# CLINICAL STUDY PROTOCOL

Evaluation of the Safety and Efficacy of Silmitasertib (CX-4945) in Combination with Standard of Care (SOC) for Treating Patients with Community-Acquired Pneumonia (CAP) Associated with SARS-CoV-2 and Influenza Viral Infections

**Protocol Number:** 

CX-4945-011

**Investigational Product:** 

Silmitasertib (CX-4945)

Phase:

2

Sponsor:

Senhwa Biosciences, Inc.

10F, No. 225, Sec. 3, Peihsin Rd., Hsintien Dist., New Taipei

City 23143, Taiwan

**Protocol Date:** 

16 August, 2024

**Protocol Version:** 

3.0

### CONFIDENTIAL

This protocol may not be reproduced or communicated to a third party without the written permission of Senhwa Biosciences, Inc.

Senhwa Biosciences, Inc. Protocol No.: CX-4945-011


Version: 3.0/ Date: 16 August, 2024

### SIGNATURE PAGE

Study Title:

Evaluation of the Safety and Efficacy of Silmitasertib (CX-4945) in Combination with Standard of Care (SOC) for Treating Patients with Community-Acquired Pneumonia (CAP) Associated with SARS-CoV-2 and Influenza Viral Infections

Objective:

Clinical Study Protocol

I have read the protocol and agree to conduct this clinical study in accordance with all stipulations of the protocol, with applicable law and regulations and in accordance with the ethical principles outlined in the Declaration of Helsinki.

SPONSOR:

Senhwa Biosciences, Inc.

Date


## PROTOCOL ACKNOWLEDGEMENT FORM

SPONSOR:

Senhwa Biosciences, Inc.

CLINICAL PROTOCOL RECEIPT

PROTOCOL NUMBER:

CX-4945-011

PROTOCOL TITLE:

Evaluation of the Safety and Efficacy of Silmitasertib (CX-4945) in Combination with Standard of Care (SOC) for Treating Patients with Community-Acquired Pneumonia (CAP) Associated with SARS-CoV-2 and Influenza Viral Infections

CONFIDENTIALITY STATEMENT:

The information contained in this document, especially unpublished data, contents and designed frameworks are the property of Senhwa Biosciences, Inc. and is therefore provided to you in confidence as a principal investigator, co-investigator, or sub-investigator, for review by you, your staffs, and an applicable Institutional Review Board (IRB) / Independent Ethics Committee (IEC). It is understood that this information will not be disclosed to others without written authorization from study sponsor.

I have received and read the Clinical (Amendment) Protocol for the above noted trial. I have agreed to conduct this clinical study in accordance with all stipulations of the protocol, with applicable law and regulations and in accordance with the ethical principles outlined in the Declaration of Helsinki

| Principal Investigator (PI) Name (print): | |
|-------------------------------------------|-------|
| Site Number: | |
| Site Name: | |
| PI Signature: | Date: |


# **SYNOPSIS**

| Title: | Combination with Standar | and Efficacy of Silmitasertib (CX-4945) in<br>d of Care (SOC) for Treating Patients with<br>amonia (CAP) Associated with SARS-CoV-2<br>ins |
|---|---|---|
| Phase: | Phase 2 | |
| Site Locations: | The study will be conducted | d in multiple centers in Taiwan. |
| Study Description and Design: | study in approximately 120 in adult outpatients with associated pneumonia. The including SARS-CoV-2 are compare the efficacy of States | enter, double-blind, randomized, interventional subjects to evaluate clinical benefit of CX-4945 SARS-CoV-2 and influenza viral infections subjects will be recruited into two domains, and influenza virus domains. The study will endard of Care (SOC) combined with CX-4945 placebo, utilizing a 1:1 allocation ratio in each ll be listed below: |
| | Domain I: SARS-Co | V-2 domain |
| | Arm 1: CX-4945 (46 | 00 mg BID for 5 days) + SOC |
| | Arm 2: Placebo + So | OC |
| | Domain II: Influenza | virus domain |
| | Arm 3: CX-4945 (4 | 00 mg BID for 5 days) + SOC |
| | Arm 4: Placebo + So | OC |
| | specified tests to determine ligible subjects who fulfi randomized into each of the | ct health information and perform protocol-<br>ne patients' eligibility. After screening visit,<br>Il all selection criteria for enrollment will be<br>arms. The CX-4945 will be administered at 400<br>s will be followed up until Day 29. |
| | 1, screening), Visit 2 (D treatment), Visit 3 (Day 7 ± follow-up), and Visit 5 (Da hospitalization and emerger influenza infection, chest X for SpO <sub>2</sub> /FiO <sub>2</sub> ratio will be a the reduction of viral present only). Safety issues, include | cs site for 5 designated visits: Visit 1 (Day $-2 \sim$ Pay 1, baseline, randomization, the start of 1, the end of treatment), Visit 4 (Day $15 \pm 2$ , $1^{st}$ by $29 \pm 3$ , $2^{nd}$ follow-up, the end of study). The next visit due to CAP related to SARS-CoV-2 or ray, body temperature, pulse oxygen saturation monitored. RT-PCR will be performed to assess tence and to measure viral load (SARS-CoV-2 ling 12-lead ECG, laboratory tests, vital signs, evaluated after treatments during study period. |
| Purpose: | The purpose of this trial is to investigate whether intervention with Silmitasertib (CX-4945) prevents the progression of CAP and moderates the elevated cytokine release associated with SARS-CoV-2 and influenza virus infection. | |
| Primary Objective | Primary Objective | Primary Endpoint |
| and Endpoints: | To evaluate the effect of intervention with | The percentage of subjects requiring hospitalization, emergency room visits, |

| | Silmitasertib (CX-4945) in addition to SOC, compared to placebo plus SOC, in preventing the progression of CAP associated with SARS-CoV-2 and influenza virus infection | or resulting in death due to progression of CAP related to SARS-CoV-2 or influenza. (Time Frame: Day 1 to Day 29) |
|---|---|---|
| Secondary Objectives and Endpoints: | Secondary Objectives To evaluate the effect of intervention with Silmitasertib (CX-4945) in addition to SOC, compared with placebo plus SOC, in enhancing the subject's clinical condition | <ul> <li>The percentage of subjects with all cause hospitalization, emergency room visits, or death during study period (Time Frame: Day 1 to Day 29)</li> <li>The percentage of subjects with improved pulmonary X-ray findings for pneumonia, relative to baseline or showing a return to normalcy (Time Frame: Baseline to Day 7, 15, and 29)</li> <li>Time to symptom resolution for fever The symptom resolution for fever is defined as body temperature lower than the following definition for 24 hours (ear temperature &lt; 38 °C, base of the tongue temperature &lt; 37.5 °C, or axillary temperature &lt; 37 °C)</li> <li>Change from baseline in SpO<sub>2</sub>/FiO<sub>2</sub> ratio (Time Frame: Day 1 to Day 7, 15, and 29)</li> <li>The percentage of subjects exhibiting disease progression is defined as an increase of score on the National Institute of Allergy and Infectious Diseases (NIAID) 8-point ordinal scale (Time Frame: Day 1 to Day 7, 15, and 29)</li> <li>The percentage of subjects exhibiting health improvement in health status Health improvement is defined as a reduction of score on the NIAID 8-point ordinal scale. (Time Frame: Day 1 to Day 7, 15, and</li> </ul> |
| | To evaluate the effect of intervention with Silmitasertib (CX-4945) in addition to SOC, compared with placebo | The percentage of subjects with a negative RT-PCR result for the SARS-CoV-2 (only for SARS-CoV-2 domain) or the influenza virus (only for influenza virus domain) on |


| | To evaluate the safety | Day 7 FilmArray data (Negative/Positive) obtained from Protocol v.1.0 will be integrated into and considered equivalent to the results for RT- PCR. (Time Frame: Day 1 to Day 7) Change from baseline in viral load in nasal secretions by RT-PCR (only for SARS-CoV-2 domain) (Time Frame: Day 1 to Day 7) Change from baseline in Ct values (only for SARS-CoV-2 domain) (Time Frame: Day 1 to Day 7) TEAEs and SAEs (Time Frame: Day 1 to Day 20) |
|---|---|---|
| | and tolerability of<br>Silmitasertib (CX-4945) | <ul> <li>(Time Frame: Day 1 to Day 29)</li> <li>Laboratory test (Time Frame: Day 1 to Day 29)</li> <li>Vital signs (Time Frame: Day 1 to Day 29)</li> <li>Electrocardiogram (ECG) results (Time Frame: Baseline to Day 29)</li> </ul> |
| Exploratory | Exploratory Objectives | Exploratory Endpoints |
| Objectives and Endpoints: | To evaluate the effect of intervention with Silmitasertib (CX-4945) in addition to SOC, compared with placebo plus SOC, on inflammatory status | Ievels on Day 7 This statistical analysis will only be conducted in subjects levels exceed the upper limit of normal (ULN) at Visit 2. (Time Frame: Day 7) Change from baseline in (Time Frame: Day 1 to Day 7, 15, and 29) Note: If the flow cytometry analyses are not performed at the local site lab, the related endpoint can be omitted. |
| | To evaluate the effect of intervention with Silmitasertib (CX-4945) | Changes from baseline in serum cytokine levels: |

| | in addition to SOC, compared with placebo plus SOC, on moderating the elevated cytokine release associated with SARS-CoV-2 and influenza virus infection (Time Frame: Day 1 to Day 7, 15, and 29) |
|---|---|
| Participant | Domain I: SARS-CoV-2 domain |
| Group/Arm: | Arm 1: CX-4945 (400 mg BID for 5 days) + SOC |
| | Arm 2: Placebo + SOC |
| | Note: The SOC within the SARS-CoV-2 domain is defined as the medications in use at each respective site for the treatment of CAP related to SARS-CoV-2 infection. |
| | Domain II: Influenza virus domain |
| | Arm 3: CX-4945 (400 mg BID for 5 days) + SOC |
| | Arm 4: Placebo + SOC |
| | Note: The SOC within the influenza virus domain is defined as the medications in use at each respective site for the treatment of CAP related to influenza virus infection. |
| Study Duration: | The study duration for each subject is up to 34 days, including screening, a treatment period of 5 days and a follow-up phase lasting until Day 29. |
| Eligibility Criteria: | Inclusion Criteria |
| | Not currently hospitalized |
| | 2. Males or females aged ≥ 18 years at the time of signing the informed consent form (ICF) |
| | 3. Patients diagnosed with viral pneumonia, as determined by the investigator, who exhibit any of the subsequent criteria: presence of respiratory symptoms or fever (ear temperature ≥ 38 °C, base of the tongue temperature ≥ 37.5 °C, or axillary temperature ≥ 37 °C) |
| | 4. With a pneumonia severity index (PSI) of risk class II or III |
| | <ol> <li>Oxygen saturation measured by pulse oximetry (SpO<sub>2</sub>) ≥ 94% on<br/>room air at sea level</li> </ol> |
| | 6. Positive test for SARS-CoV-2 or influenza virus infection, confirmed by rapid diagnostic test (excluding cases where both SARS-CoV-2 and influenza virus are positive) |
| | 7. Confirmed lower respiratory tract infection by X-ray |
| | 8. At screening, subjects capable of childbearing must provide a negative serum or urine pregnancy test. These subjects must also commit to adhering to the study-specified contraceptive methods throughout the study duration |
| | Notes: Acceptable contraceptive methods include: |


- Established use of oral, injected or implanted hormonal methods of contraception


- Placement of an intrauterine device (IUD) or intrauterine system (IUS)
- Barrier methods of contraception: condom or occlusive cap (diaphragm or cervical/vault caps)
- 9. The participant (or legal representative) agrees and is able to adhere to study protocol-stated requirements, instructions, and restrictions in the investigator's judgement. Furthermore, the participant is capable of understanding and has signed the IRB-approved Informed Consent Form (ICF)
- 10. With at least two of the risk factors listed below:

Age  $\geq$  50 years-old; cancer and a life expectancy of  $\geq$  6 months; HIV infection; immunocompromised patient; congestive heart failure (CHF), or coronary artery disease (CAD), or cardiomyopathies; chronic kidney disease (CKD); chronic liver disease; chronic lung disease; diabetes mellitus (DM); body mass index (BMI)  $\geq$  25 kg/m²; asthma; cerebrovascular disease; cystic fibrosis; dementia; or current and former smoker

## **Exclusion Criteria**

- 1. Subject received investigational treatment within 30 days prior to the study, or concurrent use of another investigational drug
- 2. Subject has a history of severe renal disease (required phosphate binders or dialysis)
- 3. Subject has chronic diarrhea, characterized by three or more loose stools daily for a minimum of four weeks
- 4. High likelihood of mortality within the next 48 hours, as assessed by the investigator
- 5. Subject showing signs of respiratory failure and mechanical ventilation is required
- 6. Subject with liver cirrhosis
- 7. Subject with hepatitis B and/or hepatitis C disease, unless the subject has an aspartate aminotransferase (AST) level ranging from 8 to 31 U/L and an alanine aminotransferase (ALT) level from 0 to 41 U/L
- 8. Known active tuberculosis
- 9. Current documented bacterial infection
- 10. Subject has a documented anaphylactic reaction, regardless of cause
- 11. Subject who has taken an antiviral agent against respiratory viral infection for a continuous duration of more than 24 hours before screening
- 12. Subject is with active gastrointestinal diseases including gastritis,


ulcerative colitis, Crohn's disease, or hemorrhagic coloproctitis 13. Subjects received warfarin within 14 days prior to screening or intend to during the screening or treatment phase 14. History of allergic reactions to any of the ingredients or components used in the manufacture of CX-4945 15. Women who are pregnant or breastfeeding, or planning pregnancy during the study **Note:** Men and women of reproductive potential must commit to effective contraception methods or abstinence during the study. Any resulting pregnancies or suspected pregnancies must be reported to the treating physician immediately. 16. ALT or AST levels > 5 times upper limit of normal (ULN) 17. eGFR <30 mL/min/1.73m<sup>2</sup> (calculated by the MDRD formula) 18. Absolute neutrophil count (ANC) <1000/μL 19. Have received treatment with a SARS-CoV-2 specific monoclonal antibody 20. Have received convalescent COVID-19 plasma treatment 21. Concurrent use of baricitinib 22. Any physical findings or illness history that may compromise study results or increase patient risk, as determined by the investigator **Treatment Regime** CX-4945 will be administered at 400 mg BID for 5 consecutive days and Duration starting on Day 1 in addition to SOC. Sample Size To ensure 120 evaluable participants (= modified Per-Protocol population) Determination and accounting for a 10% attrition rate, approximately 136 subjects will be enrolled for the study. Note that the sample size for this exploratory study is not determined by statistical power considerations, but is considered adequate for the preliminary assessment of the study's objectives. To have an adequate efficacy profile of the intervention with CX-4945 in SARS-CoV-2 and influenza virus infection, the minimum evaluable size per arm in each study domain will be 20 participants. Statistics 1. Primary hypothesis: Not applicable. 2. Efficacy population: ITT PP Other: mPP Safety population: **I**ITT **P**P Other: The Intent-to-Treat (ITT) population is defined as all randomized subjects who receive at least one dose of CX-4945 or placebo. This population will be used as the primary analysis population for efficacy endpoints and safety evaluation. The Per-Protocol (PP) population is defined as the set of subjects who (1) meet the ITT population requirements, (2) receive 80 - 120% of 10 doses of investigational product during Days 1 - 6 or die before Day 6, and (3) are not associated with any major protocol violations that have impact on

efficacy evaluation. This population will be identified before the database lock. This population will be used as the supportive analysis population for efficacy endpoints and adverse events.

The modified Per-Protocol (mPP) population is defined as the set of subjects who (1) meet the ITT population requirements, (2) receive 80 – 120% of 10 doses of investigational product during Days 1 – 6 or die before Day 6, (3) complete the required visits by Visit 4 or die before Visit 4, and (4) are not associated with any major protocol violations that have impact on efficacy evaluation by Visit 4. This population will be identified before the database lock and will be used as the supportive analysis population for efficacy endpoints.

## 3. Statistical method(s) for efficacy/safety evaluations

## General Consideration

Statistical analyses will be performed using SAS® for Windows, version 9.4 or later. All available data will be displayed via subject data listings, and summarized for each evaluation time point as appropriate by study domain (including domain-pooled) and study arm. The categorical data will be summarized with the number of subjects and percentage. Continuous data will be summarized by descriptive statistics (i.e., number of subjects, mean, standard deviation, minimum, maximum, and median). For by visit (by Day) analyses, the acceptable window for each visit will be defined in the Statistical Analysis Plan (SAP).

In general, categorical data will be analyzed by using Logistic regression (on efficacy data), Fisher's exact test or Cochran-Mantel-Haenszel test stratified by domain for comparing overall treatment group difference (treatment odds ratio for Logistic regression). For by-domain subgroup analysis on efficacy data, categorical data will be tested by using Fisher's exact test or Chi-square test.

Continuous data will be analyzed by using analysis of variance (ANOVA) on baseline data, and by using analysis of covariance (ANCOVA) on change data for comparing overall treatment group difference. Non-parametric method shall be adapted or log-transformation may be needed for non-normally distributed data. For by-domain subgroup analysis on efficacy data, continuous data will be tested by using two-sample t test or Wilcoxon Rank-sum test.

For the ANOVA, ANCOVA model and Logistic regression, factors of treatment, domain (as appropriate), site and baseline value (for post-baseline data) and other baseline factors (for post-baseline efficacy data, to be defined in the SAP, as appropriate) will be included in the model if significant, those non-statistically significant factors except treatment will be removed from the model (alpha=0.1 for interaction, 0.05 for others). The Logistic regression result will be presented with treatment odds ratio and its 95% confidence interval (CI).

All statistical tests will be two-sided and evaluated at the 0.05 level of significance. All confidence intervals, if provided, will be the 95% CI.

The most recent value before first dose administration will be defined as the baseline value; therefore, the baseline value will be the outcome of the

closest evaluation performed before or equal to the first dosing date.

### Efficacy evaluation

The primary efficacy endpoint is the percentage of subjects with the event of requiring hospitalization, emergency room visits, or resulting in death due to progression of CAP related to SARS-CoV-2 or influenza. For subjects terminated the study that event observation stopped before Day 29 and no event is observed, the subjects will be counted as 'Treatment Fail'.


The primary endpoint will be summarized in number of subjects and percentage with corresponding Clopper-Pearson exact 95% CI, and will be analyzed by using Logistic regression. Fisher's exact test or Cochran-Mantel-Haenszel test will be applied if Logistic regression is not applicable. In addition, 95% CI of treatment difference in event rate will be presented in normal approximation. Event rate including Treatment Fail rate will be tested additionally for sensitivity analysis defined in SAP.

### **Safety Evaluation**

All safety assessments, including TEAEs, physical examination, laboratory tests, vital signs, and electrocardiogram results, where indicated, will be presented using descriptive statistics.

4. Planned interim analysis: ☐Yes ■No

## SCHEDULE OF ASSESSMENTS

| Procedure/Assessments | Screening<br>Visit [15] | T | reatment Phas | e | Follow-Up | | Unscheduled<br>Visit [17] |
|---|---|---|---|---|---|---|---|
| Visit | 1 | 2 | | 3 | 4 | 5 | |
| Day | Day -2 ~ 1 | Day 1<br>(Baseline) | Day 2 ~<br>Day 6 | Day 7<br>(EOT) | Day 15 | Day 29<br>(ET/EOS) | |
| Window Period (Day) | | | | ± 1 | ± 2 | ± 3 | NA |
| Informed Consent [1] | X | | | | | | |
| Eligibility Evaluation | X | | | | | | |
| Pneumonia severity index | X | | | | | | |
| Rapid diagnostic test [12] | X | | | | | | |
| Subject<br>Demographics | X | | | | | | |
| Medical History [2] | X | X | | | | | |
| Physical Examination<br>(including body weight<br>and height) [3] | X | X | | X | X | X | Per<br>investigator's |
| Vital Signs [4] | X | X | | X | X | X | decision |
| Assessment of health<br>status using the NIAID<br>8-point ordinal scale [5] | X | X | | X | X | X | |
| Pulse Oxygen Saturation<br>for SpO <sub>2</sub> /FiO <sub>2</sub> ratio | X | X | | X | X | X | |
| 12-lead ECG | X [16] | | | X | X | X | |
| Chest X-ray | X [16] | | | X | X | X | |
| Laboratory Tests: | | | | | | | |
| Hematology [6] | X | X | | X | X | X | |
| Blood Chemistry [7] | X | X | | X | X | X | |
| Coagulation [8] | X | X | | X | X | X | |
| Serum/Urine<br>Pregnancy Test [9] | Х | | | X | | X [9#] | |
| Urinalysis [10] | X | X | | X | X | X | |
| Biomarker evaluations [11] | | X | | X | X | X | |
| RT-PCR [12] | | X | | X | | X [12#] | |
| Randomization | | X | | | | | |
| CX-4945/Placebo<br>Administration | | X [13]<br>400 mg BID | X [13]<br>400 mg BID | | | | |
| Dispense study drug | | X | | | | | X [18] |
| Return un-used drug | | | | X | | | X [18] |
| ePRO [14] | | X | X | X | X | X | |
| SOC/Supportive care | | | 9 | X (as n | eeded) | 41 | |
| Mortality Status | | X | X | X | X | X | X |
| Hospitalization events | | X | X | X | X | X | X |

Medications
Adverse Events


X

X

| Procedure/Assessments | Screening<br>Visit [15] | Ti | Treatment Phase | | se Follo | | Unscheduled<br>Visit [17] |
|---|---|---|---|---|---|---|---|
| Visit | 1 | 2 | | 3 | 4 | 5 | |
| Day | Day -2 ~ 1 | Day 1<br>(Baseline) | Day 2 ~<br>Day 6 | Day 7<br>(EOT) | Day 15 | Day 29<br>(ET/EOS) | 3.0 |
| Window Period (Day) | | | | ±1 | ± 2 | ± 3 | NA |
| Concomitant | X | X | X | X | X | X | X |

**Abbreviations**: BID = bis in die, twice a day; ECG = Electrocardiogram; EOT = end of treatment; ET = early termination; EOS = end of study; ePRO = electronic Patient Reported Outcomes;  $FiO_2 = fraction$  of inspired oxygen; SpO2 = saturation of peripheral oxygen; NA = not applicable.

X

X

X

X

- [1] Informed consent must be obtained prior to patient participation in any protocol-related activities that are not part of routine care. The results obtained from the routine care and associated tests performed within 24 hours before signing informed consent may be collected and utilized as Visit 1 data in this study (Protocol No. CX-4945-011). Additionally, body temperature measurements that fully meet protocol requirements but are taken within 24 hours before signing informed consent can be collected.
- [2] Medical history and current therapies (medications and procedures) will be included up to 2 weeks prior to screening visit. Any pre-treatment medical events will be recorded as medical history.
- [3] A complete physical exam will be performed. Height and weight should be recorded at screening visit (Visit 1) only.
- [4] Vital signs, including blood pressure, pulse rate, respiration rate, and body temperature, will be evaluated at each clinic visit. In addition, subjects will self-report their body temperature by using ePRO [14] from Day 1 to Day 7 or beyond, as needed, with the temperature being measured four times daily at 4 to 6-hour intervals.
- [5] Assessment of health status using the NIAID 8-point ordinal scale will be conducted on Screening, Days 1, 7, 15, and 29.
- [6] Hematology: hemoglobin (Hb), hematocrit (Hct), red blood cells (RBC), white blood cells (WBC), differential of leukocytes, absolute neutrophil count (ANC) and platelets.
- [7] Blood Chemistry:
  - Hepatic function indicators: total bilirubin, alkaline phosphatase (ALP), aspartate aminotransferase (AST), alanine aminotransferase (ALT), total protein, albumin
  - Renal function indicators: blood urea nitrogen (BUN), serum creatinine, and estimated Glomerular filtration rate (eGFR)
  - Electrolytes: sodium, potassium, chloride, total calcium and bicarbonate
- [8] Coagulation: Prothrombin time (PT) and international normalized ratio (INR)
- [9] ONLY performed on women of childbearing potential. # ONLY performed when early termination occurs before the completion of Visit 3.
- [10] Urinalysis: color, appearance, specific gravity, pH, protein, glucose, occult blood, ketones, leukocyte esterase, nitrite, bilirubin, urobilinogen, and microscopic examination of urine sediment.

| Evaluated biomarkers will include: |
|------------------------------------|

- [12] Swabs will be used for rapid diagnostic test, RT-PCR for presence of viral RNA (qualitative tests), Ct value and viral load:
  - At Screening, perform a rapid diagnostic test for SARS-CoV-2 or influenza virus infection using a nasopharyngeal specimen.
  - Nasopharyngeal swab for RT-PCR should be collected on Day 1 and Day 7.
  - # ONLY performed when early termination occurs before the completion of Visit 3.


Version: 3.0/ Date: 16 August, 2024 CONFIDENTIAL

- [13] Baseline assessments (on Day 1) should be conducted prior to administering the first dose of CX-4945 or placebo. Drug administration is twice daily for 5 consecutive days, starting on Day 1 and completing on Day 5, or on Day 6 if only one dose is administered on Day 1.
- [14] Patients will be instructed on the use of the Electronic Patient Reported Outcomes (ePRO) for all dose administrations and body temperature record [4] at Visit 2. Site staff will check the completeness of ePRO at Visit 3 and Visit 4, and if necessary, at Visit 5. Patients may record dose administration on Day 1  $\sim$  Day 6 and body temperature on Day 1  $\sim$ Day 7 or beyond, as needed.
- [15] Visit 1 and Visit 2 could be the same day. When Visit 1 and Visit 2 occur on the same day, the same assessments from Visit 2 can be omitted.
- [16] The results acquired from Visit 1 should serve as the baseline for the Chest X-ray and 12-lead ECG.
- [17] Adverse events, concomitant medications and hospitalization events will be recorded at an unscheduled visit (UV); other assessments will be performed at the investigator's discretion.
- [18] If the subjects have lost IPs, only one more dispensation of the investigational product is allowed per subject based on the pharmacy manual.

## TABLE OF CONTENTS

| SIG | SNATURE PAGE | . 2 |
|-----|-------------------------------------------------------|------|
| PR | OTOCOL ACKNOWLEDGEMENT FORM | . 3 |
| SYI | NOPSIS | . 4 |
| SCI | HEDULE OF ASSESSMENTS | . 12 |
| TA) | BLE OF CONTENTS | . 15 |
| | List of Tables | . 18 |
| LIS | T OF ABBREVIATIONS | |
| 1. | INTRODUCTION | . 21 |
| | 1.1. Introduction for Silmitasertib (CX-4945) | . 22 |
| | 1.2. Clinical Experience | . 23 |
| | 1.2.1. COVID-19 studies | . 23 |
| | 1.2.2. Cholangiocarcinoma study | . 24 |
| | 1.3. Study Rationale | . 25 |
| 2. | STUDY OBJECTIVES & ENDPOINTS | . 26 |
| | 2.1. Primary Objective and Endpoint | . 26 |
| | 2.2. Secondary Objective and Endpoint | . 26 |
| | 2.3. Exploratory Objectives and Endpoints | . 28 |
| 3. | STUDY DESIGN | . 29 |
| | 3.1. Overall Study Design | . 29 |
| | 3.2. Study Population | . 29 |
| | 3.2.1. Subject number | . 29 |
| | 3.2.2. Inclusion criteria | . 30 |
| | 3.2.3. Exclusion criteria | . 31 |
| | 3.3. Screen failure | . 32 |
| | 3.4. Discontinuation of Study Intervention | . 33 |
| | 3.5. Discontinuation/Withdrawal from the Study | . 33 |
| | 3.6. Method of Assigning Subjects to Treatment Groups | . 34 |
| | 3.7. Blinding | . 34 |
| | 3.8. Concomitant Therapy | . 35 |
| 4. | TREATMENTS | 36 |
| | 4.1. Detail of Study Medication | . 36 |
| | 4.1.1. Active drug | 36 |
| | 4.1.2. Placebo drug | . 36 |
| | 4.2. Dosage and Administration | . 37 |

| | 4.3. Packaging and Labeling |
|---|---|
| | 4.4. Handling and Storage |
| | 4.5. Supplies and Accountability |
| | 4.6. Treatment Compliance |
| 5. | STUDY CONDUCT |
| | 5.1. Visit Schedule |
| | 5.1.1. Visit 1 – Screening Visit (Day -2 ~ 1) |
| | 5.1.2. Visit 2 (Day 1) – Baseline, randomization, the first day of treatment |
| | 5.1.3. Visit 3 (Day $7 \pm 1$ Day) – The end of treatment (EOT) |
| | 5.1.4. Visit 4 (Day $15 \pm 2$ Days) – $1^{st}$ Follow-up |
| | 5.1.5. Visit 5 (Day 29 ± 3 Days) – 2 <sup>nd</sup> Follow-up, the end of study (EOS)/early termination (ET) |
| | 5.2. Study Assessments |
| | 5.2.1. Eligibility and informed consent |
| | 5.2.2. Demographic data, medical history, and concomitant medication |
| | 5.2.3. Pneumonia severity index |
| | 5.2.4. Efficacy Assessments |
| | 5.2.5. Safety Assessments |
| 6. | ADVERSE EVENTS |
| | 6.1. Adverse Event (AE) |
| | 6.1.1. Treatment Emergent Adverse Event (TEAE) |
| | 6.2. Serious Adverse Event (SAE) |
| | 6.3. Severity of Adverse Events |
| | 6.4. Associated with the Use of the Medication |
| | 6.5. Reporting Procedure |
| | 6.5.1. Adverse Event (AE) |
| | 6.5.2. Serious Adverse Event (SAE) |
| | 6.5.3. Pregnancy reporting |
| 7. | STATISTICAL METHODS |
| | 7.1. Sample Size Calculation |
| | 7.2. Datasets Analyzed |
| | 7.2.1. Intent-to-Treat (ITT) Population |
| | 7.2.2. Per-Protocol (PP) Population |
| | 7.2.3. Modified Per-Protocol (mPP) Population |
| | 7.3 General Consideration 57 |

| | 7.4. I | Patient Disposition | 57 |
|-----|---------|--------------------------------------------------------|----|
| | 7.5. ( | Concomitant Medications/Therapies/Medical Procedures | 8 |
| | 7.6. I | Demographic and Other Baseline Characteristics | 8 |
| | 7.7. I | Efficacy Evaluation5 | 8 |
| | 7 | 7.7.1. Analysis of Primary Efficacy Endpoint | 8 |
| | 7 | 7.7.2. Analysis of Secondary Efficacy Endpoints | 8 |
| | 7 | 7.7.3. Analysis of Exploratory Endpoint | 0 |
| | 7.8. \$ | Safety Evaluation6 | 1 |
| | 7 | 7.8.1. Treatment-emergent Adverse Events (TEAEs) | 1 |
| | 7 | 7.8.2. Physical Examination6 | 52 |
| | 7 | 7.8.3. Laboratory Tests | 2 |
| | 7 | 7.8.4. Vital Signs | 52 |
| | 7 | 7.8.5. ECG6 | 2 |
| | 7.9. I | Handling of Missing Data6 | 2 |
| 8. | DAT | A MANAGEMENT6 | 3 |
| | 8.1. I | Data Quality Assurance and Quality Control6 | 3 |
| | 8.2. I | Data Collection and Management Responsibilities | 3 |
| 9. | DIRE | ECT ACCESS TO SOURCE DATA/DOCUMENTS6 | 5 |
| | 9.1. 8 | Study Monitoring6 | 5 |
| | 9.2. A | Audits and Inspections6 | 5 |
| | 9.3. I | nstitutional Review Board/Independent Ethics Committee | 6 |
| 10. | ETHI | ICAL AND LEGAL ASPECTS6 | 7 |
| | 10.1. | Good Clinical Practice | 7 |
| | 10.2. | Delegation of Investigator Responsibilities | 7 |
| | 10.3. | Subject Information and Informed Consent | 7 |
| | 10.4. | Subject Rights and Confidentiality | 8 |
| | 1 | 0.4.1. Subject confidentiality | 8 |
| | 1 | 0.4.2. Study discontinuation | 8 |
| | 10.5. | Protocol Amendments | 8 |
| | 10.6. | Approval of the Study Protocol and Amendments | 8 |
| | 10.7. | Publication policy6 | 9 |
| | Protoc | col Amendment History | 0 |
| 11 | DEFE | PDENCES | 2 |

### Senhwa Biosciences, Inc. Protocol No.: CX-4945-011

### CONFIDENTIAL


## **List of Tables**

| Table 5-1 PSI Algorithm | 43 |
|---|---|
| Table 5-2 Discharge from hospital (Outpatients Subsequently Hospitalized) | 45 |
| Table 5-3 NIAID 8-point ordinal scale | 46 |
| Table 6-1 Grading scales of AEs | 52 |
| Table 6-2 Causality categories between AEs and study drug | 53 |

# LIST OF ABBREVIATIONS

| Abbreviations | Terms and Definitions |
|---|---|
| ADL | Activities of daily living |
| ADR | Adverse drug reaction |
| AE | Adverse Event |
| ALT | Alanine Aminotransferase |
| ANC | Absolute neutrophil count |
| ANCOVA | Analysis of Covariance |
| AST | Aspartate Aminotransferase |
| AUC | Area Under Curve |
| ATC | Anatomic Therapeutic Classification |
| BUN | Blood urea nitrogen |
| CAD | Coronary artery disease |
| CAP | Community-Acquired Pneumonia |
| CARDS | Acute respiratory distress syndrome |
| CHF | Congestive heart failure |
| CI | Confidence interval |
| CK2 | Casein kinase II |
| CKD | Chronic kidney disease |
| CRA | Clinical Research Associate |
| CRF | Case Report Form |
| CRO | Contract Research Organization |
| Ct | Cycle threshold value |
| CTCAE | Common Terminology Criteria for Adverse Events |
| DM | Diabetes mellitus |
| ECF | Extended care facility |
| ECG | Electrocardiography |
| ECMO | Extracorporeal membrane oxygenation |
| EDC | Electronic data capture |
| eGFR | Estimated Glomerular filtration rate |
| ePRO | Electronic Patient Reported Outcome |
| EOS | End Of Study |
| EOT | End of treatment |
| ET | Early termination |
| FAS | Full Analysis Set |
| FiO <sub>2</sub> | Fraction of Inspired Oxygen |
| GCP | Good Clinical Practice |
| HB | Hemoglobin |
| Hct | Hematocrit |
| HEENT | Head, ears, eyes, nose, throat |
| ICH | International Council for Harmonisation of Technical Requirements for |
| | Pharmaceuticals for Human Use |
| ICU | Intensive care unit |
| ID | Identification |
| IEC | Independent Ethics Committee |

| Abbreviations | Terms and Definitions |
|---------------|-------------------------------------------------------|
| 9300 | |
| INR | International normalized ratio |
| IP | Investigational product |
| IRB | Institutional Review Board |
| ITT | Intent-to-Treat |
| LDH | lactate dehydrogenase |
| LOCF | Last Observation Carry Forward |
| MedDRA | Medical Dictionary for Regulatory Activities |
| mTOR | Mechanistic target of rapamycin |
| NCS | No clinical significance |
| NLR | Neutrophil to lymphocyte ratio |
| NIAID | National Institute of Allergy and Infectious Diseases |
| PLR | Platelet-to-lymphocyte ratio |
| PPS | Per Protocol Set |
| PRO | Patient Reported Outcome |
| PSI | Pneumonia Severity Index |
| PT | Prothrombin time |
| QD | Quaque die |
| RBC | Red blood cells |
| RT-PCR | Reverse transcription polymerase chain reaction |
| SAE | Serious Adverse Event |
| SAF | Safety population |
| SHH | Sonic Hedgehog |
| $SpO_2$ | Saturation of Peripheral Oxygen |
| STAT3 | Signal transducer and activator of transcription 3 |
| SUSAR | Suspected Unexpected Serious Adverse Reaction |
| TEAE | Treatment emergent adverse events |
| TESAE | Treatment-emergent serious adverse event |
| TFDA | Taiwan Food and Drug Administration |
| <b>建造建</b> 装基 | |
| ULN | Upper limit of normal |
| WBC | White blood cells |


### 1. INTRODUCTION

Community-acquired pneumonia (CAP) is a serious clinical problem which refers to an acute infection of the pulmonary parenchyma acquired outside of the hospital. The worldwide incidence of community-acquired pneumonia varies between 1.5 to 14 cases per 1000 person-years. The mortality rate is as high as 6% for hospitalized patients and 23% for patients admitted to the intensive care unit. The elderly adults ≥ 65 years-old with comorbidities have a higher risk of CAP, with a 2% hospitalization rate. In WHO 2020 report, 15% of children <5 years of age die from pneumonia. Moreover, immunocompromised patients have also an increased risk in CAP than general population. Lifestyle factors also affect the risk factors of CAP, including smoking, high alcohol consumption, being underweight, poor oral hygiene and frequent contact with children. <sup>1,2,3</sup>


The clinical presentation of CAP varies, ranging from mild symptoms that are fever, chills, cough productive of purulent sputum, dyspnea, pleuritic chest pain, and weight loss to severe symptoms that characterized by respiratory distress and sepsis.<sup>1,2</sup> In elder patients, more frequently symptoms present in confusion or worsening of pre-existing conditions, and without chest signs or fever.<sup>4</sup>

The cause of CAP could be a range of bacteria and virus. The most frequently detected pathogens in patients with CAP is *Streptococcus pneumoniae* (pneumococcus, about 30% to 35% of cases in the US and Europe <sup>4</sup>) and respiratory viruses (around 22% cases<sup>5</sup>). However, the microbial etiology of CAP could not be detected in ~50% of patients due to the failure to obtain an adequate culture sample before the initiation of therapy, and the inconsistent availability of newly improved molecular tests.

Viral pneumonia is common in the very young and in the elderly patients, while a steep decline in the incidence of viral pneumonia was observed from adolescence to 50~60 years-old patients, except people with immunosuppression. However, the epidemiological condition varies by pandemic season and region, such as flu epidemics or coronavirus disease 2019 (COVID-19) pandemics. Viral pneumonia generally occurs in 3 kinds of mechanisms: (1) viral particles would inoculate directly into the lung (e.g., respiratory syncytial virus (RSV) or influenza); (2) virus spread in a contiguous fashion from viral infection to upper respiratory tract (e.g., measles); and (3) hematogenous spread from a distant viral infection (e.g., cytomegalovirus). Sometimes, viral respiratory tract infections could lead to primary viral pneumonias and also predispose to secondary bacterial pneumonias. The availability of PCR-based multiplex tests enables the simultaneous identification of a wide number of viruses in viral pneumonia diagnosis. At least 26 viruses associated with CAP have now been identified that most pronounced is influenza virus infection. RSV is the predominant viral pathogen in the severe CAP. And a meta-analysis study in 2016 wrote by M Burk *et al.* for CAP patient associated with viral infection

Protocol No.: CX-4945-011

by using PCR identification, 31 researches (10762 subjects) were included. Of these researches, 24.5% (95% confidence interval (CI): 21.5-27.5%) patients have viral infection, 10% (95% CI: 8-11%) patients were revealed dual bacterial and viral infection. The most common identified viruses were influenza (8%), followed by rhinovirus (5.7%), coronavirus (3.3%), and respiratory syncytial virus (2.2%). There was no statistical significance among viral infection in short-term mortality, but the odds of death were significantly higher compared with patients without dual infection (OR: 2.1, 95% CI: 1.32-3.31; p=0.002; I<sup>2</sup> =0%).8 In the recent year, ongoing outbreak of COVID-19 is reporting high mortality and morbidity in the world. People from all age groups are susceptible to SARS-CoV-2; however, the proportion of SARS-CoV-2 infection in children is lower than that of adults. Severe COVID-19 pneumonia is a huge challenge in clinical management. 9 For people hospitalized with covid-19, 15-30% will go on to develop covid-19 associated acute respiratory distress syndrome (CARDS) that they require ventilatory support. 10

### 1.1. Introduction for Silmitasertib (CX-4945)

CX-4945 is a first-in-class potent and highly selective small molecule inhibitor of casein kinase II (CK2) that interacts competitively with the ATP-binding site of CK2 subunit alpha, leading towards the inhibition of several downstream signaling pathways. CK2 is involved in regulation of signaling through protein pathways phosphorylation and also plays a multifunctional role in signal transduction, transcriptional control, apoptosis and inflammation. Overexpression of CK2 was observed in diseases with high proliferative activities, inflammatory reaction and dysregulated immune response (viral infections, auto-immune inflammations, cancer).

The biological activity of CX-4945 has been evaluated in both in vitro and in vivo studies:

- CX-4945 demonstrated strong anti-viral efficacy in human cells infected by SARS-CoV-2 (pre-clinical in vitro study)11
- CX-4945 significantly reduced replication of human papillomavirus in vivo<sup>12</sup>
- In several pre-clinical and clinical trials in the diseases driven by pro-inflammatory cytokines CX-4945 demonstrated ability to significantly reduce plasma level of interleukins (IL-6, IL-8, IL-17) in vitro and in vivo (inflammatory breast cancer, Alzheimer's disease, autoimmune encephalomyelitis). 13
- CK2 inhibitor down-regulated replication, budding and release of influenza virus in preclinical studies<sup>14</sup>

- CK2 inhibitor reduced phosphorylation dependent ICP27 protein export, which is necessary for its ability to export herpes simplex viral RNAs<sup>15</sup>
- CX-4945 also demonstrated anti-tumor activity in a variety of primary human xenografts and tumor cell line xenograft models and in clinical trials

### 1.2. Clinical Experience

#### 1.2.1. COVID-19 studies

CX-4945 may potentially quell virus-provoked aberrant hyperactivation of the innate immune system by inhibition of upregulated CK2 protein kinase, preferentially restoring normal host cell cytokine regulation, and attenuating viral replication in patients with COVID-19 infection, thereby preventing disease progression and improving clinical outcomes.

CX-4945 was used for COVID-19 treatment in a phase I dose selection study (Protocol number: CX4945-AV04-phase I) and a phase II study (Protocol number: CX4945-AV01-IIT) under IND 152726.

In the phase I study, 30 healthy subjects were randomized into 200mg QD, 200mg BID, and 400mg BID cohorts, respectively, with 1:1:1 allocation. The total duration of the treatment was 5 days. Subjects were followed up on Day 14 after the start of the treatment. A total of 7 TEAEs in 7 subjects (23.33%) were reported as drug-related TEAEs. The most common drug-related TEAEs were diarrhea in 5 subjects in 400mg BID cohort and 1 subject in 200mg BID cohort. All of the drug-related TEAEs were mild. During study period, no treatment-emergent serious adverse event (TESAE) or death was reported. In clinical laboratory evaluations, vital signs, physical examinations, and 12-lead ECGs evaluations, no clinical significant finding was observed. Therefore, all dosing regimens (200mg QD, 200mg BID, or 400mg BID) were safe and well-tolerated. 16

In the phase II study, a randomized, multi-center, two-arm parallel-group controlled interventional prospective study in subjects with moderate COVID-19 was conducted. Total 20 outpatient subjects were enrolled and randomized in a 1:1 ratio in two groups, including 10 subjects in CX-4945 in combination with SOC and 10 subjects in SOC only. CX-4945 1000 mg BID for 14 days was applied. In terms of COVID-19 history, mean (SD) duration of the 20 subjects were 2.8 (2.24) days with mean symptom duration of 6.3 (2.95) days. None of these subjects had COVID-19 vaccination history. In the safety results, five subjects suffered treatment related AEs in CX-4945 group, but none of these AEs were equal or greater than Grade 3. Only 2 subjects experienced SAEs and 3 subjects underwent Grade ≥ 3 AEs in the study, but all of which were drug-unrelated. Neither death nor Suspected Unexpected Serious Adverse Reaction (SUSAR) was reported through the study. Several clinical

significant laboratory values were detected, and most of them returned to normal or no clinical significance (NCS).<sup>17</sup>

With respective to time to clinical signs normalization, subjects in CX-4945 group had a median time of 7 (95% CI: $1.0 \sim .$ ) compared to SOC group of 11 (95% CI: $5.0 \sim 16.0$ ). With regard to time to COVID-19-related symptom recovery, subjects receiving CX-4945 had a median time of 7 (95% CI: $4.0 \sim 12.0$ ) compared to 14 (95% CI: $7.0 \sim .$ ) of SOC group. In terms of time to oxygen saturation level normalization, subjects in CX-4945 group had a mean time of 1 compared to SOC group of 1 (95% CI: $1.0 \sim 5.0$ ). In terms of investigation of clinical benefit by EQ-D5-5L and NIAID 8-Point Clinical Progression Outcomes Scale, no significant difference was found between the two groups. No significant difference was detected on viral load and viral clearance proportion between two groups except for Day 8. Regarding changes in inflammatory markers, almost all results of two treatment groups were normal or NCS except for some due to medical history or AEs. 17

## 1.2.2. Cholangiocarcinoma study

CX-4945 is currently under development in several oncology programs in adults and in children with recurrent/advanced or metastatic cancer. CX-4945 is used as an antitumor agent that inhibits the Sonic Hedgehog signaling pathway (basal cell carcinoma, medulloblastoma) and/or DNA repair in tumor cells damaged by chemotherapy (cholangiocarcinoma) through inhibition of CK2.

Several phase I and II clinical trials of CX-4945 in cancer patients have been completed to date (e.g., solid tumors, multiple myeloma, and cholangiocarcinoma), and there is one ongoing phase I study (basal cell carcinoma; protocol number: CX-4945-07) under IND 102181 and one ongoing phase II studies (medulloblastoma; protocol number: PBTC-053) under IND 137563.

In a phase 1b/2 study (Protocol number: S4-13-001) under the US IND 144857, the subjects received CX-4945 1000 mg BID for 10 days with gemcitabine and cisplatin (G+C) on Days 1 and 8 of a 21-day cycle (n =55) or gemcitabine and cisplatin only (n =29). The median PFS was 11.2 months (95% CI, 7.6, 14.7) in CX-4945 with G+C group and 5.8 months (95% CI, 3.1, not evaluable [NE]) (p = 0.0496) in G+C only group. The median overall survival was 17.4 months (95% CI, 13.4, 25.7) in CX-4945 with G+C group versus 14.9 months (95% CI, 9.9, NE) in G+C only group. The overall response rate and disease control rate was 34.0% versus 30.8%, 86.0% versus 88.5% with CX-4945 with G+C versus G+C only groups, respectively. The most common TEAEs (all grades) with CX-4945/G+C versus G+C were diarrhea (70% versus 13%), nausea (59% vs. 30%), fatigue (47% vs. 47%), vomiting (39% vs. 7%), and anemia (39% vs. 30%). <sup>18</sup>

### 1.3. Study Rationale

| Silmitasertib (CX-4945) is an inhibitor of the protein kinase CK2 (CK2, also known as casein kinas |
|---|
| 2). It exhibits both antiviral and anti-inflammatory properties against COVID-19 in vitro, and |
| showcasing its potential to improve the time to clinical signs normalization and time to COVID-19 |
| related symptom recovery (CX4945-AV01-IIT; US IND 152726). CK2 modulates inflammator |
| pathways, including CK2 by CX-494. |
| diminishes the secretion of |
| stimulated with NiSO4 (Bourayne |
| et al., 2017). <sup>20</sup> Hence, CX-4945 offers potential against viral infections and may moderate the elevated |
| cytokine release during inflammation. We aim to further investigate the safety and efficacy o |
| Silmitasertib (CX-4945) in combination with standard of care (SOC) for treating patients with |
| community-acquired pneumonia (CAP) associated with SARS-CoV-2 and influenza viral infections. |

This is a Phase II multi-center, double-blind, randomized, interventional study in approximately 120 subjects to evaluate clinical benefit of CX-4945 in adult outpatients with SARS-CoV-2 and influenza viral infection-associated pneumonia. The study will compare the efficacy of SOC combined with CX-4945 against SOC paired with a placebo, utilizing a 1:1 allocation ratio. CX-4945 will be administered at 400 mg BID for up to 5 days. This dose derives from one completed Phase I studies wherein healthy volunteers were administered CX-4945 at increment doses of 200 mg QD, 200 mg BID and 400 mg BID over a span of 5 days. The purpose of this trial is to investigate whether intervention with Silmitasertib (CX-4945) prevents the progression of CAP and moderates the elevated cytokine release associated with SARS-CoV-2 and influenza virus infection.


2. Study Objectives & Endpoints

# 2.1. Primary Objective and Endpoint

| Primary Objective | Primary Endpoint |
|---|---|
| To evaluate the effect of intervention with Silmitasertib (CX-4945) in addition to SOC, compared to placebo plus SOC, in preventing the progression of CAP associated with SARS-CoV-2 and influenza virus infection | The percentage of subjects requiring hospitalization, emergency room visits, or resulting in death due to progression of CAP related to SARS-CoV-2 or influenza. (Time Frame: Day 1 to Day 29) |

# 2.2. Secondary Objective and Endpoint

| Secondary Objectives | Secondary Endpoints |
|---|---|
| To evaluate the effect of intervention with Silmitasertib (CX-4945) in addition to SOC, compared with placebo plus SOC, in enhancing the subject's clinical condition | <ul> <li>The percentage of subjects with all cause hospitalization, emergency room visits, or death during study period (Time Frame: Day 1 to Day 29)</li> <li>The percentage of subjects with improved pulmonary X-ray findings for pneumonia, relative to baseline or showing a return to normalcy (Time Frame: Baseline to Day 7, 15, and 29)</li> <li>Time to symptom resolution for fever The symptom resolution for fever will be defined as body temperature lower than the following definition for 24 hours (ear temperature &lt; 38°C, base of the tongue temperature &lt; 37.5°C, or axillary temperature &lt; 37°C)</li> <li>Change from baseline in SpO<sub>2</sub>/FiO<sub>2</sub> ratio (Time Frame: Day 1 to Day 7, 15, and 29)</li> <li>The percentage of subjects exhibiting disease progression in health status</li> <li>Disease progression is defined as an increase of score on the</li> </ul> |

| Secondary Objectives | Secondary Endpoints |
|---|---|
| | National Institute of Allergy and Infectious Diseases (NIAID) 8-point ordinal scale. (Time Frame: Day 1 to Day 7, 15, and 29) • The percentage of subjects exhibiting health improvement in health status Health improvement is defined as a reduction of score on the NIAID 8-point ordinal scale. (Time Frame: Day 1 to Day 7, 15, and 29) |
| To evaluate the effect of intervention with Silmitasertib (CX-4945) in addition to SOC, compared with placebo plus SOC, on reducing viral presence | <ul> <li>The percentage of subjects with a negative RT-PCR result for the SARS-CoV-2 (only for SARS-CoV-2 domain) or the influenza virus (only for influenza virus domain) on Day 7 FilmArray data (Negative/Positive) obtained from Protocol v.1.0 will be integrated into and considered equivalent to the results for RT-PCR. (Time Frame: Day 1 to Day 7)</li> <li>Change from baseline in viral load in nasal secretions by RT-PCR (only for SARS-CoV-2 domain) (Time Frame: Day 1 to Day 7)</li> <li>Change from baseline in Ct values (only for SARS-CoV-2 domain) (Time Frame: Day 1 to Day 7)</li> </ul> |
| To evaluate the safety and tolerability of Silmitasertib (CX-4945) | <ul> <li>TEAEs and SAEs (Time Frame: Day 1 to Day 29)</li> <li>Laboratory test (Time Frame: Day 1 to Day 29)</li> <li>Vital signs (Time Frame: Day 1 to Day 29)</li> <li>Electrocardiogram (ECG) results (Time Frame: Baseline to Day 29)</li> </ul> |

# 2.3. Exploratory Objectives and Endpoints

| <b>Exploratory Objectives</b> | Exploratory Endpoints |
|---|---|
| To evaluate the effect of intervention with Silmitasertib (CX-4945) in addition to SOC, compared with placebo plus SOC, on inflammatory status | <ul> <li>The percentage of subjects achieving normalized levels on Day 7 This statistical analysis will only be conducted in subjects whose levels exceed the upper limit of normal (ULN) at Visit 2. (Time Frame: Day 7)</li> <li>Change from baseline in Change from baseline in levels exceed the upper limit of normal (ULN) at Visit 2. (Time Frame: Day 7)</li> <li>Change from baseline in levels exceed the upper limit of normal (ULN) at Visit 2. (Time Frame: Day 7)</li> <li>And 29)</li> <li>Note: If the flow cytometry analyses for levels are not performed at the local site lab, the related endpoint be omitted.</li> </ul> |
| To evaluate the effect of intervention with Silmitasertib (CX-4945) in addition to SOC, compared with placebo plus SOC, on moderating the elevated cytokine release associated with SARS-CoV-2 and Influenza virus infection | Changes from baseline in serum cytokine levels: Cytokines to be quantified; (Time Frame: Day 1 to Day 7, 15, and 29) |


### 3. STUDY DESIGN

### 3.1. Overall Study Design

This is a Phase II, multi-center, double-blind, randomized, interventional study in approximately 120 subjects to evaluate clinical benefit of CX-4945 in adult outpatients with SARS-CoV-2 and influenza viral infection-associated pneumonia. The subjects will be recruited into two domains, including SARS-CoV-2 and Influenza virus domains. The study will compare the efficacy of SOC combined with CX-4945 against SOC paired with a placebo, utilizing a 1:1 allocation ratio in each domain. The study arms will be listed below:

### Domain I: SARS-CoV-2 domain

Arm 1: CX-4945 (400 mg BID for 5 days) + SOC

Arm 2: Placebo + SOC

#### Domain II: Influenza virus domain

Arm 3: CX-4945 (400 mg BID for 5 days) + SOC

Arm 4: Placebo + SOC

Screening visit will collect health information and perform protocol-specified tests to determine patients' eligibility. After screening visit, eligible subjects who fulfill all selection criteria for enrollment will be randomized into each of the arms. The CX-4945 will be administered at 400 mg BID for 5 days. Subjects will be followed up until Day 29.

Subjects will return to clinics site for 5 designated visits: Visit 1 (Day -2~1, screening), Visit 2 (Day 1, baseline, randomization, the start of treatment), Visit 3 (Day 7 ± 1, the end of treatment), Visit 4 (Day 15 ± 2, 1<sup>st</sup> follow-up), and Visit 5 (Day 29 ± 3, 2<sup>nd</sup> follow-up, the end of study). The hospitalization and emergency visit due to CAP related to SARS-CoV-2 or influenza infection, chest X-ray, body temperature, pulse oxygen saturation for SpO<sub>2</sub>/FiO<sub>2</sub> ratio will be monitored. RT-PCR will be performed to assess the reduction of viral presence and to measure viral load (SARS-CoV-2 only). Safety issues, including 12-lead ECG, laboratory test, vital signs, and adverse events will be evaluated after treatments during study period.

### 3.2. Study Population

### 3.2.1. Subject number

A total of 120 evaluable subjects (= modified Per-Protocol population) will be enrolled into the study.

The subjects in each domain will be randomized with 1:1 allocation ratio into active drug plus SOC arm and placebo plus SOC arm. The study arms will be as the following:

### Domain I: SARS-CoV-2 domain

Arm 1: CX-4945 (400 mg BID for 5 days) + SOC

Arm 2: Placebo + SOC

Note: The SOC within the SARS-CoV-2 domain is defined as the medications in use at each respective site for the treatment of CAP related to SARS-CoV-2 infection.

#### Domain II: Influenza virus domain

Arm 3: CX-4945 (400 mg BID for 5 days) + SOC

Arm 4: Placebo + SOC

Note: The SOC within the influenza virus domain is defined as the medications in use at each respective site for the treatment of CAP related to influenza virus infection.

### 3.2.2. Inclusion criteria

Subjects meeting all of the following criteria will be considered for enrollment into the study:

- 1. Not currently hospitalized
- 2. Males or females aged  $\geq$  18 years at the time of signing the informed consent form (ICF)
- 3. Patients diagnosed with viral pneumonia, as determined by the investigator, who exhibit any of the subsequent criteria: presence of respiratory symptoms or fever (ear temperature ≥ 38 °C, base of the tongue temperature ≥ 37.5 °C, or axillary temperature ≥ 37 °C)
- 4. With a pneumonia severity index (PSI) of risk class II or III
- 5. Oxygen saturation measured by pulse oximetry (SpO₂) ≥94% on room air at sea level
- 6. Positive test for SARS-CoV-2 or influenza virus infection, confirmed by rapid diagnostic test (excluding cases where both SARS-CoV-2 and influenza virus are positive)
- 7. Confirmed lower respiratory tract infection by X-ray
- 8. At screening, subjects capable of childbearing must provide a negative serum or urine pregnancy test. These subjects must also commit to adhering to the study-specified contraceptive methods throughout the study duration

Notes: Acceptable contraceptive methods include:

- Established use of oral, injected or implanted hormonal methods of contraception
- Placement of an intrauterine device (IUD) or intrauterine system (IUS)
- Barrier methods of contraception: condom or occlusive cap (diaphragm or cervical/vault caps)
- 9. The participant (or legal representative) agrees and is able to adhere to study protocol-stated requirements, instructions, and restrictions in the investigator's judgement. Furthermore, the participant is capable of understanding and has signed the IRB-approved Informed Consent Form (ICF)
- 10. With at least two of the risk factors listed below:

Age  $\geq$  50 years-old; cancer and a life expectancy of  $\geq$  6 months; HIV infection; immunocompromised patient; congestive heart failure (CHF), or coronary artery disease (CAD), or cardiomyopathies; chronic kidney disease (CKD); chronic liver disease; chronic lung disease; diabetes mellitus (DM); body mass index (BMI)  $\geq$  25 kg/m<sup>2</sup>; asthma; cerebrovascular disease; cystic fibrosis; dementia; or current and former smoker

### 3.2.3. Exclusion criteria

- Subject received investigational treatment within 30 days prior to the study, or concurrent use of another investigational drug
- 2. Subject has a history of severe renal disease (required phosphate binders or dialysis)
- Subject has chronic diarrhea, characterized by three or more loose stools daily for a minimum of four weeks
- 4. High likelihood of mortality within the next 48 hours, as assessed by the investigator
- 5. Subject showing signs of respiratory failure and mechanical ventilation is required
- 6. Subject with liver cirrhosis
- 7. Subject with hepatitis B and/or hepatitis C disease, unless the subject has an aspartate aminotransferase (AST) level ranging from 8 to 31 U/L and an alanine aminotransferase (ALT) level from 0 to 41 U/L
- 8. Known active tuberculosis
- 9. Current documented bacterial infection
- 10. Subject has a documented anaphylactic reaction, regardless of cause

- 11. Subject who has taken an antiviral agent against respiratory viral infection for a continuous duration of more than 24 hours before screening
- 12. Subject is with active gastrointestinal diseases including gastritis, ulcerative colitis, Crohn's disease, or hemorrhagic coloproctitis
- 13. Subjects received warfarin within 14 days prior to screening or intend to during the screening or treatment phase
- History of allergic reactions to any of the ingredients or components used in the manufacture of CX-4945
- 15. Women who are pregnant or breastfeeding, or planning pregnancy during the study
  Note: Men and women of reproductive potential must commit to effective contraception methods

or abstinence during the study. Any resulting pregnancies or suspected pregnancies must be reported to the treating physician immediately.

- 16. ALT or AST levels > 5 times upper limit of normal (ULN)
- 17.  $eGFR < 30 \text{ mL/min}/1.73\text{m}^2$  (calculated by the MDRD formula)
- 18. Absolute neutrophil count (ANC) <1000/μL
- 19. Have received treatment with a SARS-CoV-2 specific monoclonal antibody
- 20. Have received convalescent COVID-19 plasma treatment
- 21. Concurrent use of baricitinib
- 22. Any physical findings or illness history that may compromise study results or increase patient risk, as determined by the investigator.

### 3.3. Screen failure

Screen failures are defined as participants who consent to participate in the clinical study but are not subsequently enrolled in the study. A minimal set of screen failure information is required to ensure transparent reporting of screen failure participants to meet the Consolidated Standards of Reporting Trials (CONSORT) publishing requirements and to respond to queries from regulatory authorities. Minimal information includes demography, screen failure details, and eligibility criteria.

Individuals who do not meet the criteria for participation in this study (screen failure) may not be rescreened.

Protocol No.: CX-4945-011 CONFIDENTIAL Version: 3.0/ Date: 16 August, 2024

### 3.4. Discontinuation of Study Intervention

Discontinuation of study product CX-4945/placebo does not mean discontinuation from the study, and the remaining study procedures will be completed as designated by this protocol. If a clinically significant finding is identified following the initiation of study treatment, the Investigator (or designee) will determine if any change in subject management is necessary. However, a subject should be discontinued from study product CX-4945/placebo in any of the following circumstances:

- A suspected Grade 3 or higher treatment-related AE (according to Common Terminology Criteria for Adverse Events (CTCAE) version 5.0)
- Any treatment-related SAE
- A subject receives baricitinib
- A subject receives warfarin
- The subject is pregnant

## 3.5. Discontinuation/Withdrawal from the Study

Subjects will be followed and monitored over the course of the study stated in Section 5.1 Visit Schedule. If a subject does not attend any of the regularly scheduled visits, the subject will not be deemed as withdrawn, but the missed visit(s) will be considered as missing data in the study registry. Subjects may be discontinued from study product CX-4945 (Section 3.4) at the discretion of the Investigator if any severe, untoward effects occur to the subjects during the treatment phase. However, subjects may not be terminated from the study because of AEs.

If a subject, whether continuing study product CX-4945 or not, fails to return to any scheduled visits (i.e., lost to follow-up), or if the Investigator determines that it is in subject's best interest to be prematurely withdrawn from the study, the Investigator must determine the primary reason for subject's premature withdrawal and document this incidence in the eCRF, including the date of occurrence and the reason(s). All study-related information collected prior to subject's withdrawal will be retained and maintained in the study analysis unless otherwise explicitly requested by the subject; however, no further efforts will be made to obtain or record additional medical information about the subject. Subjects will be withdrawn from the study prematurely due to any of the following circumstances:

- Subject (or legal representative) decides to withdraw consent at any time.
- Subject, determined by the Investigator (or designee), is no longer physically or mentally feasible for further participation in the study.
- Subject is lost to follow-up.

• The sponsor terminates the study.

All collected/generated data and information about the subjects in the study prior to the time of study discontinuation will be recorded and analyzed, including the date and reason(s) to discontinue the study.

All subjects who have received at least one dose of study medication will be encouraged to complete all tests scheduled for the ET wherever possible at the time of the subject's withdrawal within 7 days.

### 3.6. Method of Assigning Subjects to Treatment Groups

The study treatment will be randomly assigned to subjects. The randomized sequence of study treatments will be generated by a qualified biostatistician. The randomization schedule will be kept and maintained by the designated personnel before the study begins and until the database lock. The biostatistician prepares the schedule with a 1:1 randomization ratio (CX-4945: Placebo) by stratified randomization with study domains and study sites strata. Also, block permutation is used for generating randomization schedule. Eligible subjects will receive a random number at randomization. The subject will receive the corresponding treatment assigned by the EDC system. For any reason that a subject withdraws from the study prematurely after the randomization, his/her randomization number will not be reused. The next eligible subject will receive the lowest available randomization number.

### 3.7. Blinding

This is a double-blind study. Neither the subject nor the investigators, clinic administrators, or sponsor staff who involve in the treatment or clinical evaluation of the subjects will be aware of the treatment received either at the time of randomization or later, throughout the conduct of the trial. Assigned unblinded team may include study site stuff, CRO's personnel and/or Senhwa Biosciences, Inc's personnel. Other personnels involved in the study (the investigator and the clinical monitor) will be blinded until the database lock.

The treatment codes will not be prematurely broken unless an emergency situation, when the appropriate management of the subject necessitated acknowledgement of the treatment allocation, occurred. In the event of a medical emergency, if possible, the medical monitor should be contacted first to discuss the need for unblinding. For unblinding a subject, the treatment code blind can be obtained by the investigator, by accessing the EDC system.

The sponsor must be notified immediately if the treatment code blind is broken.

## 3.8. Concomitant Therapy

- 1. The following medication should be prohibited during the specified period:
  - (1) Warfarin is prohibited 14 days prior to screening and the treatment phase.
  - (2) Any other investigational treatment within 30 days before Screening and during study
- 2. The routine use of antibiotics is not recommended. Antibiotics may be used if bacterial infections are present or suspected. The type of antibiotic will be selected based on the subject's clinical disease status and symptoms with discretion of investigator.


## 4. TREATMENTS

# 4.1. Detail of Study Medication

## 4.1.1. Active drug

| Study medication | CX-4945 |
|---|---|
| Characteristics & Physical State | The isolated CX-4945 Sodium Salt is pale yellow to yellow solid which is formulated in an opaque blue, shell-gelatin capsule. |
| Dose(s) | 200 mg/capsule |
| Dosage and Frequency | CX-4945 will be administered at 400 mg BID for 5 consecutive days starting on Day 1 in addition to SOC. |
| Administration route | Immediate release, oral administration |
| Mechanism of Action | CX-4945 is an inhibitor of Casein Kinase II (CK2) with anti-viral and anti-inflammatory effects. It interacts competitively with the ATP-binding site of CK2 subunit alpha, leading to the inhibition of several downstream signaling pathways. |
| Pharmacological category | Antiviral Drug |
| Storage | Store at temperature between 15-30°C. |
| Manufacturer | Senhwa Biosciences, Inc. |

## 4.1.2. Placebo drug

| Study medication: | CX-4945 Placebo |
|---|---|
| Characteristics & Physical State | The placebo drug is identical in appearance to the CX-4945 with the same excipient ingredients, but without the active compound. |
| Dose(s) | 200 mg/capsule |
| Dosage and Frequency | The dosage and frequency are the same as active drug. |
| Administration route | Immediate release, oral administration |
| Storage | Store at temperature between 15-30°C. |
| Manufacturer | Senhwa Biosciences, Inc. |
4.2. Dosage and Administration

Subjects will take two capsules of 200 mg CX-4945 or placebo, along with water twice daily on an

empty stomach (preferably two hours after finishing a meal). It is recommended to take one capsule at

a time with a 10-minute interval between each capsule to avoid a clumping effect. After taking the

capsules, subjects are encouraged to avoid food intake, except for water, for at least 2 hours.

4.3. Packaging and Labeling

Packaging: CX-4945 are supplied as 200 mg strength auto-filled capsules (AFCs) in size 1, opaque

blue capsules. Seventy (70) CX-4945 capsules (or placebo) are packaged in a 120 cc wide mouth round

white HDPE bottle with a 38 mm cap with induction seal. The bottle contains a polyester coil and 1 g

Sorb-IT® desiccant. Senhwa Biosciences will arrange the preparation, packaging and distribution of

the study drugs.

Labeling: All study medication will be supplied in identical package, and the label will include the

required regulatory agency caution statements, the protocol number, the Sponsor's identification,

manufacturer's name, storage conditions, and expiry date.

4.4. Handling and Storage

The study medication will be handled by the investigator or the designated pharmacist for management

and dispensation. All supplies for this study should be kept under adequate security and storage

conditions. CX-4945 should be stored in the container provided, between 15 °C and 30 °C, as indicated

on the label, and should be protected from moisture, freezing, and bright light

4.5. Supplies and Accountability

The investigator or the pharmacist will inventory and acknowledge receipt of all shipments of study

medication. All study medication must be kept in a locked area with access restricted to designated

study personnel. The study medication must be stored in accordance with the manufacturer's

instructions. The investigator or pharmacist will also keep accurate records of the quantities of study

medication dispensed and used by each subject. The site monitor will periodically check the supplies

of study medication held by the investigator or the pharmacist to ensure accountability of all study

medication used.


# 4.6. Treatment Compliance

Site staff will dispense study medications to all subjects ensuring proper administration of the investigational product (IP). Patients will be instructed on using ePRO to keep a dosing record for all dose administrations. Patients will be instructed to bring the dosing record and all unused study medication and empty study medication containers at Visit 3. The dosing record will be reviewed and the IP will be counted, documented, and recorded by site staff. The investigator or sub-investigator will check the compliance status of each patient based on the number of prescribed IP, number of returned IP, or number of lost IP, and describe compliance status in the medical record or other source documents, as well as checking data integrity in reference to the IP inventory at each visit.

# Protocol No.: CX-4945-011 CONFIDENTIAL Version: 3.0/ Date: 16 August, 2024

# 5.1. Visit Schedule

5. STUDY CONDUCT

# 5.1.1. Visit 1 -Screening Visit (Day $-2 \sim 1$ )

After a subject has signed the informed consent document, he or she will be enrolled after screening for selection criteria. The following assessments should be evaluated at this visit:

- (1) Obtain signed informed consent
- (2) Check subject's eligibility: inclusion and exclusion criteria
- (3) Collect demographic data
- (4) Collect general medical history
- (5) Conduct physical exam: It should be also recorded a complete physical exam, height, and weight
- (6) Measure vital signs
- (7) Collect NIAID 8-point ordinal scale
- (8) Assess pulse oxygen saturation: measure SpO2 and record FiO2
- (9) Perform 12-lead ECG
- (10) Perform chest X-ray
- (11) Collect urine and blood samples for the following laboratory tests
  - Hematology
  - Blood Chemistry
  - Coagulation
  - Urinalysis
- (12) Perform pregnancy test: Only for female with child bearing potential
- (13) Record Pneumonia Severity Index (PSI) risk class
- (14) Collect nasopharyngeal swab samples for rapid diagnostic test
- (15) Collect prior and concomitant medications

#### 5.1.2. Visit 2 (Day 1) – Baseline, randomization, the first day of treatment

The following procedures should be evaluated at the visit:

- Collect any change of medical history. Any pre-treatment medical events will be recorded as medical history
- (2) Conduct physical exam

- (3) Measure vital signs
- (4) Collect NIAID 8-point ordinal scale
- (5) Assess pulse oxygen saturation: measure SpO<sub>2</sub> and record FiO<sub>2</sub>
- (6) Collect urine and blood samples for the following laboratory tests.
  - Hematology
  - Blood Chemistry
  - Coagulation
  - Urinalysis
  - Biomarker evaluations
- (7) Collect nasopharyngeal swab samples for RT-PCR
- (8) Randomization
- (9) Dispense study drug. The study drugs will be administered for 5 consecutive days starting on Day 1 and completing on Day 5, or on Day 6 if only one dose is administered on Day 1.
- (10) Provide SOC/supportive care (as needed)
- (11) Record any change of concomitant medication
- (12) Instruct the use of the Electronic Patient Reported Outcomes (ePRO) for dose administrations and body temperature record
- (13) Record hospitalization events and ER visit, if any
- (14) Check mortality status
- (15) Record adverse events after drug administration, if any

# 5.1.3. Visit 3 (Day $7 \pm 1$ Day) – The end of treatment (EOT)

The following assessments should be evaluated at this visit:

- (1) Conduct physical exam
- (2) Measure vital signs
- (3) Collect NIAID 8-point ordinal scale
- (4) Assess pulse oxygen saturation: measure SpO<sub>2</sub> and record FiO<sub>2</sub>
- (5) Perform 12-lead ECG
- (6) Perform chest X-ray
- (7) Collect urine and blood samples for the following laboratory tests.
  - Hematology
  - Blood Chemistry
  - Coagulation


- Urinalysis
- Biomarker evaluations
- (8) Perform pregnancy test: Only for female with child bearing potential
- (9) Collect nasopharyngeal swab samples for RT-PCR
- (10) Check ePRO completion status
- (11) Provide SOC/supportive care (as needed)
- (12) Check drug accountability and compliance. Return all unused study drugs and empty containers
- (13) Record hospitalization events and ER visit, if any
- (14) Record any change of concomitant medication
- (15) Record adverse events and check mortality status, if needed

# 5.1.4. Visit 4 (Day $15 \pm 2$ Days) – $1^{st}$ Follow-up

The following assessments should be evaluated at this visit:

- (1) Conduct physical exam
- (2) Measure vital signs
- (3) Collect NIAID 8-point ordinal scale
- (4) Assess pulse oxygen saturation: measure SpO<sub>2</sub> and record FiO<sub>2</sub>
- (5) Perform 12-lead ECG
- (6) Perform chest X-ray
- (7) Collect urine and blood samples for the following laboratory tests.
  - Hematology
  - Blood Chemistry
  - Coagulation
  - Urinalysis
  - · Biomarker evaluations
- (8) Provide SOC/supportive care (as needed)
- (9) Check ePRO completion status
- (10) Record hospitalization events and ER visit, if any
- (11) Record any change of concomitant medication
- (12) Record adverse events and check mortality status, if needed

# 5.1.5. Visit 5 (Day $29 \pm 3$ Days) $-2^{nd}$ Follow-up, the end of study (EOS)/early termination (ET)

The following assessments should be evaluated at this visit:

- (1) Conduct physical exam
- (2) Measure vital signs
- (3) Collect NIAID 8-point ordinal scale
- (4) Assess pulse oxygen saturation: measure SpO<sub>2</sub> and record FiO<sub>2</sub>
- (5) Perform 12-lead ECG
- (6) Perform chest X-ray
- (7) Collect urine and blood samples for the following laboratory tests.
  - Hematology
  - Blood Chemistry
  - Coagulation
  - Urinalysis
  - Biomarker evaluations
- (8) Perform pregnancy test: Only for female with child bearing potential when early termination occurs before the completion of Visit 3
- (9) Collect nasopharyngeal swab samples for RT-PCR (only performed when early termination occurs before the completion of Visit 3)
- (10) Provide SOC/supportive care (as needed)
- (11) Check ePRO completion status (as needed)
- (12) Record hospitalization events and ER visit, if any
- (13) Record any change of concomitant medication
- (14) Record adverse events and check mortality status, if needed

#### 5.2. Study Assessments

# 5.2.1. Eligibility and informed consent

Subjects will be screened prior to the start of the study treatment. All assessments will be performed after the subjects have signed and dated the informed consent form.

The investigator or a designee will explain the nature of the study to subjects. The subject will be given an informed consent form to be read carefully before agreeing to take part in the study and before the study-specific procedures take place. The informed consent form should be reviewed, signed, and dated by the subject and the investigator. A copy of the statement will be given to the subject, and the


original should be maintained by the investigator in the site master file. After informed consent being obtained, designed procedures and assessments will be initiated to determine eligibility.

### 5.2.2. Demographic data, medical history, and concomitant medication

Demographic data will be collected at the screening visit. Demographic data includes birth year, age, and sex.

Any pre-treatment medical events will be recorded as medical history. The general medical history within 2 weeks before Screening Visit should be recorded at Screening Visit. The general medical history includes chronic diseases, allergic history, surgical history, and disease of interests, such as pulmonary, gastrointestinal, cardiovascular, cerebrovascular, and autoimmune events, cystic fibrosis, dementia, and acute or chronic infection. History of severe renal disease and documented anaphylactic reaction should be recorded in a lifetime basis.

Concomitant medication will be recorded when subjects received the following:

- Medication from 2 weeks prior to screening visit to end of the study
- Any investigational treatment within 30 days prior to the study
- SARS-CoV-2 specific monoclonal antibody or convalescent COVID-19 plasma treatment prior to screening

#### 5.2.3. Pneumonia severity index

For each subject, the risk class of Pneumonia Severity Index (PSI) will be recorded. PSI is a clinical predication rule which can be used to calculate the probability of morbidity and mortality for community acquired pneumonia. It is used to predict the need for hospitalization in people with pneumonia.

Table 5-1 PSI Algorithm

| Presence of: | |
|-----------------------------------|--------|
| Over 50 years of age | Yes/No |
| Altered mental status | Yes/No |
| Pulse ≥125/minute | Yes/No |
| Respiratory rate >30/minute | Yes/No |
| Systolic blood pressure <90 mm Hg | Yes/No |
| Temperature <35 °C or ≥40 °C | Yes/No |

| History of: | |
|--------------------------|--------|
| Neoplastic disease | Yes/No |
| Congestive heart failure | Yes/No |
| Cerebrovascular disease | Yes/No |
| Renal disease | Yes/No |
| Liver disease | Yes/No |

| Demographics | Points Assigned |
|----------------------------------------------|-----------------|
| If Male | +Age (yr) |
| If Female | +Age (yr) - 10 |
| Nursing home resident | +10 |
| Comorbidity | |
| Neoplastic disease | +30 |
| Liver disease | +20 |
| Congestive heart failure | +10 |
| Cerebrovascular disease | +10 |
| Renal disease | +10 |
| Physical Exam Findings | |
| Altered mental status | +20 |
| Pulse ≥125/minute | +10 |
| Respiratory rate >30/minute | +20 |
| Systolic blood pressure <90 mm Hg | +20 |
| Temperature <35 °C or ≥40 °C | +15 |
| Lab and Radiographic Findings | |
| Arterial pH <7.35 | +30 |
| Blood urea nitrogen ≥30 mg/dl (9 mmol/liter) | +20 |
| Sodium <130 mmol/liter | +20 |
| Glucose ≥250 mg/dl (14 mmol/liter) | +10 |
| Hematocrit <30% | +10 |


| Partial pressure of arterial O <sub>2</sub> <60mmHg | +10 |
|------------------------------------------------------|-----|
| Pleural effusion | +10 |
| $\Sigma < 70 = $ Risk Class II | |
| $\Sigma 71-90 = \underline{\mathbf{Risk Class III}}$ | |
| $\Sigma$ 91-130 = Risk Class IV | |

A pneumonia severity index will be assessed at screening visit.

# 5.2.4. Efficacy Assessments

# 5.2.4.1. Hospitalization and Emergency Room Visit

If a participant is hospitalized or during emergency room (ER) visit, procedures and assessments will continue per the visit schedule. Hospitalization is defined as inpatient admission and more details are listed in **Section 5.2.5.6**. Hospitalization event will be followed up until Day 29.

This table describes discharge from hospital scenarios if an outpatient is subsequently hospitalized.

Table 5-2 Discharge from hospital (Outpatients Subsequently Hospitalized)

| If hospital discharge | Then |
|---|---|
| Occurs prior to Day 29 | Subjects will be asked to complete the remaining study assessments at the time points indicated in the visit schedule |
| Occurs on the same day as a scheduled study visit | If the scheduled study assessments are performed during hospitalization and the circumstances meet all the following criteria, assessments do not need to be repeated. • The scheduled study assessments have been performed within 8 hours of discharge. • There has been no change in clinical status. • The information is available to the site. |

# 5.2.4.2. Chest X-ray

Chest X-ray will be performed at Visits 1, 3, 4, and 5. The results obtained at Visit 1 should be baseline before the start of treatment. The findings will be evaluated by the investigators and noted as "Normal", "Abnormal, non-clinical significant (NCS)" or "Abnormal, clinical significant (CS)" with comments in the CRF/eCRF. Any clinical significant abnormal findings should be recorded as an adverse event during the study. Post-treatment pneumonia status, as assessed by the chest X-ray, will be categorized as 'Worsen', 'No Change', 'Improved' or 'Normal'.

# 5.2.4.3. National Institute of Allergy and Infectious Diseases (NIAID) 8-point ordinal scale

The NIAID 8-point ordinal scale used in this study is as follows:

Table 5-3 NIAID 8-point ordinal scale

| Score | Description |
|---|---|
| 1 | Not hospitalized with no limitation of activities |
| 2 | Not hospitalized - limitation of activities or home oxygen, or both |
| 3 | Hospitalized with no supplemental oxygen, and no ongoing medical care |
| 4 | Hospitalized with no supplemental oxygen, but with ongoing medical care |
| 5 | Hospitalized with requirement of supplemental oxygen |
| 6 | Hospitalized with need of non-invasive ventilation or high flow oxygen supplementation |
| 7 | Hospitalized with invasive mechanical ventilation or extracorporeal membrane oxygenation (ECMO) |
| 8 | Death |

Disease severity will be evaluated using the National Institute of Allergy and Infectious Diseases (NIAID) 8-point ordinal scale. Higher score indicates deterioration in the clinical status. Disease progression is defined as an increase of score on the NIAID 8-point ordinal scale, such as from Score 1 to Score 3. Health improvement is defined as a reduction of score on the NIAID 8-point ordinal scale, such as from Score 4 to Score 2.

#### 5.2.4.4. RT-PCR

Nasopharyngeal swabs will be used to perform RT-PCR for the following tests:

Presence of viral RNA (qualitative result: positive or negative)


Ct values (SARS-CoV-2 Domain only)

Viral load (SARS-CoV-2 Domain only)

Fully validated RT-PCR tests shall be performed. RT-PCR tests for SARS-CoV-2 Domain will be conducted in the central lab, while testing for the presence of viral RNA for influenza Virus Domain will be performed at each local site lab.

# 5.2.4.5. Mortality status

Mortality status will be followed up until Day 29 if applicable.

# 5.2.4.6. Electronic Patient Reported Outcome (ePRO)

An ePRO will be used for subjects to record body temperature from Day 1 to Day 7 or beyond to confirm fever-free (as Section **5.2.5.2 Vital signs**) and the IP intake from Day 1 up to Day 6.

#### 5.2.5. Safety Assessments

#### 5.2.5.1. Physical examination

A complete physical examination will be performed at every visit, including the examination of general appearance, HEENT (head, ears, eyes, nose, throat), neck (including thyroid), lymph nodes, skin, cardiovascular, pulmonary, abdomen, neurological system and musculoskeletal/joints.

A complete physical examination will be performed at each visit. Height and weight will be collected at Visit 1 (Screening Visit) only.

## 5.2.5.2. Vital signs

The pulse rate, blood pressures in sitting position, respiratory rate, and body temperature will be assessed and recorded in clinic site at each visit. The body temperature assessed at site on Day 1 should be baseline before the start of treatment. Any clinically significant abnormal findings should be record as an adverse event during the study.

After the first dose of CX-4945 or placebo administration on Day 1, subjects will self-measure their body temperature and record it in ePRO four times a day, every 4 to 6 hours.

#### To confirm fever-free:

After the temperature falls below the fever definition, the subject will continue recording for a minimum of 24 hours.

#### 5.2.5.3. Electrocardiogram

The results of ventricular rate, PR interval, QRS interval, QT interval, and RR interval will be recorded, if available. Corrected QT interval (QTc) will be calculated using Fridericia formula. ECG will be evaluated by the investigators and noted as "Normal", "Abnormal, non-clinical significant (NCS)" or "Abnormal, clinical significant (CS)" with comments in the CRF/eCRF. The test may be repeated if the original result is questionable.

#### 5.2.5.4. Pulse oxygen saturation

Measuring the amount of oxygen-carrying hemoglobin in the blood relative to the amount of hemoglobin not carrying oxygen will be performed at each visit. Pulse oxygen saturation will be measured using a standard pulse oximeter, oxygen analyzer, or physiologic monitor. Record the FiO<sub>2</sub> accompanying each SpO<sub>2</sub> measurement. Oxygen saturation to fraction of inspired oxygen ratio (SpO<sub>2</sub>/FiO<sub>2</sub>) will be calculated for statistical analyses.

# 5.2.5.5. Laboratory test

The following laboratory analyses will be performed. Reference ranges will be used by the investigator to assess the laboratory data for clinical significance and pathological changes.

#### Hematology

Hemoglobin (Hb), Hematocrit (Hct), Red Blood Cells (RBC), White Blood Cells (WBC), differential of leukocytes, Absolute Neutrophil Count (ANC) and platelets.

#### **Blood Chemistry**

- Hepatic function indicators: total bilirubin, alkaline phosphatase (ALP), aspartate
   aminotransferase (AST), alanine aminotransferase (ALT), total protein, albumin
- Renal function indicators: BUN, Serum creatinine, and eGFR
- Electrolytes: sodium, potassium, chloride, total calcium and bicarbonate

# Coagulation

Prothrombin time (PT) and International Normalized Ratio (INR)

#### Urinalysis

Color, appearance, specific gravity, pH, protein, glucose, occult blood, ketones, leukocyte esterase, nitrite, bilirubin, urobilinogen, and microscopic examination of urine sediment (including red blood cells, white blood cells, epithelial cells, bacteria, casts, and crystals.)


#### Biomarker evaluations



#### 5.2.5.6. Hospitalization events

If a subject is admitted to the hospital, the participant will remain in the study and follow the procedures outlined in the visit schedule. Hospitalization is defined as inpatient admission.

The date of hospitalization events will be recorded in the CRF and includes:

- Hospitalization
- Emergency room visit: only for dosed subjects that last 24 hours or longer will be included
- ICU admittance
- Extended care facility (ECF) admittance: ECF events will only be documented for subjects dosed in the trial who experience adverse events (AEs) and require additional medical support in the ECF, such as respiratory therapy to address the AEs. The requirement for additional medical support in the ECF is considered comparable to hospitalization as a discretion by the investigator. This means ECF events occurring before trial enrollment will not be documented. Additionally, enrolled subjects without experiencing AEs move to the ECF after enrollment will not be considered hospitalized and do not need to be entered into the EDC.
- Discharge

# 5.2.5.7. Clinical Status and Medications/Procedures of Special Interest

The subject's clinical status and concurrent medications/procedures of special interest will be recorded in the CRF, including the level of consciousness, limitation on activities due to CAP, and requirements for the following:


- Ongoing hospital medical care
- Supplemental oxygen
- Non-invasive ventilation or a high flow oxygen device
- Mechanical ventilation
- ECMO
- Additional organ support (e.g., pressors, renal replacement)

# 5.2.5.8. Respiratory Support

Once enrolled in the study, subjects may be managed with high-flow nasal cannula, noninvasive positive pressure ventilation or any other form respiratory support as needed per investigator discretion

#### 5.2.5.9. Pregnancy test

A urine or blood pregnancy test should be performed in women of childbearing potential at screening visit and Day 7. Subject should carry out efficient birth control throughout the study period.

# 5.2.5.10. Treatment Emergent Adverse Events (TEAEs)

The treatment emergent adverse events will be collected from the start of treatment to the end of study.

The detail of adverse event will be referred to **Section 6 Adverse Events**.

#### 6. ADVERSE EVENTS

The treatment emergent adverse event (TEAE) and serious adverse event (SAE) will be recorded from the start of treatment until the end of study.

Any pre-treatment medical events will be recorded as medical history.

#### 6.1. Adverse Event (AE)

An adverse event (AE) can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding, for example), symptom, or disease temporally associated with the use of a medicinal product, whether or not considered related to the study medication. (Definition per International Conference on Harmonization [ICH]). A medical occurrence fulfills the definition of SAE in section 6.2 is also an AE.

Except for SAEs, Adverse Events are NOT:

- Clinical events related to expected progression of COVID-19 or influenza.
- Medical or surgical procedures (e.g., surgery, endoscopy, tooth extraction, transfusion).
   However, the condition that leads to the procedure is an AE.
- Situations where an untoward medical occurrence has not occurred (e.g., hospitalization for elective surgery, social and/or convenience admissions).

#### 6.1.1. Treatment Emergent Adverse Event (TEAE)

A treatment-emergent adverse event (TEAE) is defined as any unfavorable and unintended disease or its sign (including an abnormal laboratory value) in a subject who received the study drug, irrespective of the causal relationship with the study drug.

#### 6.2. Serious Adverse Event (SAE)

The definition of a Serious Adverse Event (SAE) is any untoward (negative with respect to the subject's pre-operative condition) medical occurrence that:

- Results in death.
- Is life threatening (immediately as it occurred, not had it become worse at some time in the future),
- Requires hospitalization (or a prolongation of hospitalization in already hospitalized patients),
- Results in a persistent or significant disability or incapacity, or

• Is a congenital anomaly or birth defect.

There are medical events that may not require inpatient hospitalization, be immediately life threatening, or result in death but may jeopardize the subject or may require intervention to prevent one of the other outcomes listed before. Medical and scientific judgments should be exercised in deciding whether an event should be reported as a "Serious Adverse Event."

Nevertheless, the following events will NOT be reported as a SAE:

- Hospitalization due to social reasons in absence of an adverse event
- Hospitalization due to surgery or procedure planned before entry into the study (must be documented in the CRF)
- Hospitalization for elective treatment of a pre-existing condition that did not worsen from baseline

# 6.3. Severity of Adverse Events

The investigator should use clinical judgment in assessing the severity of events not directly experienced by the subject (e.g., laboratory abnormalities). The grade refers to the severity of the AE using CTCAE Version 5.0 (published on November 27, 2017). The CTCAE displays Grade 1 to 5 with unique clinical descriptions of severity for each AE as shown in below:

Table 6-1 Grading scales of AEs

| Grades of AEs | Description |
|---|---|
| Grade 1 | Mild; asymptomatic or mild symptoms; clinical or diagnostic observations |
| | only; intervention not indicated. |
| Grade 2 | Moderate; minimal, local or noninvasive intervention indicated; limiting age- |
| | appropriate instrumental ADL* |
| Grade 3 | Severe or medically significant but not immediately life-threatening |
| | hospitalization or prolongation of hospitalization indicated; disabling, limiting |
| | self-care ADL** |
| Grade 4 | Life-threatening consequences; urgent intervention indicated. |
| Grade 5 | Death related to AE. |

<sup>\*</sup> Activities of daily living (ADL) refer to preparing meals, shopping for groceries or clothes, using the telephone, managing money, etc.

<sup>\*\*</sup> Self-care ADL refer to bathing, dressing and undressing, feeding self, using the toilet, taking medication, and not bedridden.

6.4. Associated with the Use of the Medication

# rotocol No.: CX-4945-011 CONFIDENTIAL Version: 3.0/ Date: 16 August, 2024

An adverse event is considered associated with the use of the drug if the attribution is certain, probably/likely, possible, or unlikely by the definitions listed as follows. The causal relationship between AEs and study drug modified from WHO-UMC system for standardized case causality assessment.

Table 6-2 Causality categories between AEs and study drug

| Causality term | Assessment criteria |
|---|---|
| Certain | <ul> <li>Event or laboratory test abnormality, with plausible time relationship<br/>to drug intake</li> </ul> |
| | <ul> <li>Cannot be explained by disease or other drugs</li> </ul> |
| | <ul> <li>Response to withdrawal plausible (pharmacologically, pathologically)</li> </ul> |
| | Event definitive pharmacologically or phenomenologically (i.e., an objective and specific medical disorder or a recognized phenomenop) |
| | pharmacological phenomenon) |
| D-1-11-/17-1 | Rechallenge satisfactory, if necessary |
| Probable / Likely | <ul> <li>Event or laboratory test abnormality, with reasonable time relationship<br/>to drug intake</li> </ul> |
| | <ul> <li>Unlikely to be attributed to disease or other drugs</li> </ul> |
| | <ul> <li>Response to withdrawal clinically reasonable</li> </ul> |
| | Rechallenge not required |
| Possible | <ul> <li>Event or laboratory test abnormality, with reasonable time relations<br/>to drug intake</li> </ul> |
| | <ul> <li>Could also be explained by disease or other drugs</li> </ul> |
| | <ul> <li>Information on drug withdrawal may be lacking or unclear</li> </ul> |
| Unlikely | • Event or laboratory test abnormality, with a time to drug intake that makes a relationship improbable (but not impossible) |
| | Disease or other drugs provide plausible explanations |
| Unrelated | <ul> <li>Occurred before dosing</li> <li>Due wholly to factors other than study treatment</li> </ul> |

#### 6.5. Reporting Procedure

#### 6.5.1. Adverse Event (AE)

Any AE occurring from the time the subject takes the first dose of the IP will be collected as treatmentemergent adverse events (TEAE) and the safety analysis will be carried out with TEAE. All TEAEs, regardless of seriousness, severity, or presumed relationship to study regimen, will be evaluated and recorded by investigators preferably with a diagnosis or medical terminology instead of signs, symptoms, and/or other clinical information on the TEAE form of CRF until recoverable or stable without a further follow-up by investigators' opinions. All measures required for adverse event management must be recorded in the source document and reported according to sponsor instructions.

#### 6.5.2. Serious Adverse Event (SAE)

As any SAE occurs, the investigator must inform sponsor or its delegate within 24 hours of their knowledge of the event by email, fax or telephone.

It is the responsibility of Investigators to review all documents (e.g., site progress notes, laboratory, and diagnostics reports) relative to the AEs/SAEs/SUSARs and record on the appropriate documents. Investigator will transmit the related copies of patient's medical records for SUSAR cases to sponsor. In this instance, all patient identifiers will be blinded on the copies of the medical records prior to submission to the sponsor ASAP. The sponsor should file the initial report of SUSAR to FDA/TFDA within 15 days (7 days for death or life-threatening events) after aware of the event. Completed follow-up report for death or life-threatening events must be filed within 15 days and/or till recoverable or stable without a further follow-up by investigators' opinions.

The SAE and SUSAR shall be reported promptly according to the reporting procedure of each IRB(s).

# 6.5.3. Pregnancy reporting

Any subject and subject's female partner who becomes pregnant during the study period should be recorded and the information regarding this pregnancy should be collected. When a subject suspects a pregnancy during the study period, a pregnancy test should be conducted. Once pregnancy is confirmed, the subject should be withdrawn from the study (Section 3.5). The pregnancy should be reported to the sponsor using the pregnancy report form. The Obstetrician/Gynecologist of the female subject or male subject's partner should be notified the study information. Because information of specific tests regarding this IP is not clear yet, whenever possible, a pregnancy should be followed to term or to any premature terminations reported. Additionally, the status of the mother and child should

be reported to the sponsor after delivery. Although pregnancy occurring during the study is not considered as an adverse event, abnormal pregnancy outcomes (e.g., spontaneous abortion, fetal death, stillbirth, congenital anomalies, and ectopic pregnancy) are consider SAEs.

# 7. STATISTICAL METHODS

# 7.1. Sample Size Calculation

To ensure 120 evaluable participants (Section 3.2.1) and accounting for a 10% attrition rate, approximately 136 subjects will be enrolled for the study. Note that the sample size for this exploratory study is not determined by statistical power considerations, but is considered adequate for the preliminary assessment of the study's objectives. To have an adequate efficacy profile of the intervention with CX-4945 in SARS-CoV-2 and influenza virus infection, the minimum evaluable size per arm in each study domain will be 20 participants.

# 7.2. Datasets Analyzed

# 7.2.1. Intent-to-Treat (ITT) Population

The ITT population is defined as all randomized subjects who receive at least one dose of CX-4945 or placebo. This population will be used as the primary analysis population for efficacy endpoints and the analysis population for baseline data, safety and exploratory endpoints.

# 7.2.2. Per-Protocol (PP) Population

The PP population is defined as the set of subjects who meet the ITT population and below requirements:

- Receive 80 120% of 10 doses of the IP during Days 1 6 or die before Day 6
- · Not associated with any major protocol violations that have impact on efficacy evaluation

This population will be identified before the database lock and will be used as the supportive analysis population for efficacy endpoints and AE.

#### 7.2.3. Modified Per-Protocol (mPP) Population

The mPP population is defined as the set of subjects who meet the ITT population and below requirements:

- Receive 80 120% of 10 doses of the IP during Days 1 6 or die before Day 6
- Complete the required visits by Visit 4 or die before Visit 4
- Not associated with any major protocol violations that have impact on efficacy evaluation by Visit

This population will be identified before the database lock and will be used as the supportive analysis population for efficacy endpoints.

#### 7.3. General Consideration

Statistical analyses will be performed using SAS® for Windows, version 9.4 or later. All available data will be displayed via subject data listings, and summarized for each evaluation time point as appropriate by study domain (including domain-pooled) and study arm. The categorical data will be summarized with the number of subjects and percentage. Continuous data will be summarized by descriptive statistics (i.e., number of subjects, mean, standard deviation, minimum, maximum, and median). For by visit (by Day) analyses, the acceptable window for each visit will be defined in the Statistical Analysis Plan (SAP).

In general, categorical data will be analyzed by using Logistic regression (on efficacy data), Fisher's exact test or Cochran-Mantel-Haenszel test stratified by domain for comparing overall treatment group difference (treatment odds ratio for Logistic regression). For by-domain subgroup analysis on efficacy data, categorical data will be tested by using Fisher's exact test or Chi-square test.

Continuous data will be analyzed by using analysis of variance (ANOVA) on baseline data, and by using analysis of covariance (ANCOVA) on change data for comparing overall treatment group difference. Non-parametric method shall be adapted or log-transformation may be needed for non-normally distributed data. For by-domain subgroup analysis on efficacy data, continuous data will be tested by using two-sample t test or Wilcoxon Rank-sum test.

For the ANOVA, ANCOVA model and Logistic regression, factors of treatment, domain (as appropriate), site and baseline value (for post-baseline data) and other baseline factors (for post-baseline efficacy data, to be defined in the SAP, as appropriate) will be included in the model if significant, those non-statistically significant factors except treatment will be removed from the model (alpha=0.1 for interaction, 0.05 for others). The Logistic regression result will be presented with treatment odds ratio and its 95% confidence interval (CI).

All statistical tests will be two-sided and evaluated at the 0.05 level of significance. All confidence intervals, if provided, will be the 95% CI.

The most recent value before first dose administration will be defined as the baseline value; therefore, the baseline value will be the outcome of the closest evaluation performed before or equal to the first dosing date.

#### 7.4. Patient Disposition

The disposition of all patients who signed an ICF will be provided. The number of subjects screened, screen failed, randomized, received at least one treatment, completed, and discontinued during the

study, as well as the reasons for all discontinuations will be summarized.

#### 7.5. Concomitant Medications/Therapies/Medical Procedures

All medications will be coded to matching Anatomic Therapeutic Classification (ATC) codes using the most recent version of the WHO Drug Dictionary. Percentage of taking prior medication and concomitant medications will be presented, respectively, by the highest ATC level.

All medical procedures including surgery will be coded using the most recent version of Medical Dictionary for Regulatory Activities (MedDRA). Percentage of receiving prior medical procedures and concomitant medical procedures will be presented, respectively, by the system organ class and preferred term.

All coding terms will be included in the subject data listing.

#### 7.6. Demographic and Other Baseline Characteristics

Demographics and baseline characteristics including medical history, prior and concomitant medications/therapies and treatment exposure up to Day 6 and total treatment exposure will be summarized using appropriate statistics mentioned in section 7.3.

#### 7.7. Efficacy Evaluation

# 7.7.1. Analysis of Primary Efficacy Endpoint

The primary efficacy endpoint is the percentage of subjects with the event of requiring hospitalization, emergency room visits, or resulting in death due to progression of CAP related to SARS-CoV-2 or influenza. For subjects terminated the study that event observation stopped before Day 29 and no event is observed, the subjects will be counted as 'Treatment Fail'.

The primary endpoint will be summarized in number of subjects and percentage with corresponding Clopper-Pearson exact 95% CI, and will be analyzed by using Logistic regression. Fisher's exact test or Cochran-Mantel-Haenszel test will be applied if Logistic regression is not applicable. In addition, 95% CI of treatment difference in event rate will be presented in normal approximation. Event rate including Treatment Fail rate will be tested additionally for sensitivity analysis defined in SAP.

#### 7.7.2. Analysis of Secondary Efficacy Endpoints

The percentage of subjects with all cause hospitalization, emergency room visit or death during study period


This endpoint will be analyzed in the same way as on primary endpoint.

# The percentage of subjects with improved pulmonary X-ray findings for pneumonia, relative to baseline or showing a return to normalcy


Pneumonia status will be tabulated descriptively by visit. Percentage of 'Improved' or 'Normal' will be presented with the corresponding Clopper-Pearson exact 95% CI, and tested by using Fisher's exact test or Cochran-Mantel-Haenszel test.

## Time to symptom resolution for fever

Fever (ear temperature  $\geq$  38°C, base of the tongue temperature  $\geq$  37.5°C, or axillary temperature  $\geq$  37°C) status will be tabulated descriptively by visit. For subgroup of subjects with fever at baseline, time to symptom resolution for fever will be analyzed by using Log-rank test stratified by domain, and step plot of Kaplan-Meier graph will be provided. For subjects without symptom resolution for fever, censoring at (1) the last temperature measurement time point of the subject, (2) the last temperature measurement time point of all subjects, will both be derived for analysis.

## Change from baseline in SpO<sub>2</sub>/FiO<sub>2</sub> ratio

The SpO<sub>2</sub>/FiO<sub>2</sub> ratio and changes in SpO<sub>2</sub>/FiO<sub>2</sub> ratio will be summarized descriptively by visit. The change from baseline will be analyzed by using ANCOVA.

# The percentage of subjects exhibiting disease progression / health improvement in health status

NIAID score and changes in NIAID score will be tabulated descriptively by visit. For protocol version 1.0, 6-Point Ordinal Scale collected for subjects of Influenza Virus domain will be converted to corresponding NIAID score using table below and combined with NIAID score for analyses.

| 6-point | 6-point Ordinal Scale | NIAID 8- | NIAID 8-point Description |
|---|---|---|---|
| Score | Description | point Score | |
| 1 | Death | 8 | Death |
| 2 | In the intensive care unit (ICU) Plus condition: with invasive mechanical ventilation or extracorporeal membrane oxygenation (ECMO) | 7 | Hospitalized with invasive mechanical ventilation or extracorporeal membrane oxygenation (ECMO) |
| 2 | In the intensive care unit (ICU) Plus condition: with non-invasive ventilation or high flow oxygen supplementation | 6 | Hospitalized with need of non-invasive ventilation or high flow oxygen supplementation |
| 2 | In the intensive care unit (ICU) Plus condition: with supplemental oxygen | 5 | Hospitalized with requirement of supplemental oxygen |
| 2 | In the intensive care unit (ICU) Plus condition: with no supplemental oxygen, but with ongoing Standard of Care | 4 | Hospitalized with no supplemental oxygen, but with ongoing medical care |
| 3 | Non-ICU hospitalization, requiring supplemental oxygen Plus condition: with invasive mechanical ventilation or extracorporeal membrane oxygenation (ECMO) | 7 | Hospitalized with invasive mechanical ventilation or extracorporeal membrane oxygenation (ECMO) |

| 6-point<br>Score | 6-point Ordinal Scale Description | NIAID 8-<br>point Score | NIAID 8-point Description |
|---|---|---|---|
| 3 | Non-ICU hospitalization, requiring supplemental oxygen Plus condition: with non-invasive ventilation or high flow oxygen supplementation | 6 | Hospitalized with need of non-invasive ventilation or high flow oxygen supplementation |
| 3 | Non-ICU hospitalization, requiring supplemental oxygen Plus condition: with supplemental oxygen | 5 | Hospitalized with requirement of supplemental oxygen |
| 4 | Non-ICU hospitalization, not requiring supplemental oxygen Plus condition: with ongoing Standard of Care | 4 | Hospitalized with no supplemental oxygen, but with ongoing medical care |
| 4 | Non-ICU hospitalization, not requiring supplemental oxygen <u>Plus condition: without no ongoing Standard of Care</u> | 3 | Hospitalized with no supplemental oxygen, and no ongoing medical care |
| 5 | Not hospitalized, but unable to resume normal activities | 2 | Not hospitalized - limitation of activities or home oxygen, or both |
| 6 | Not hospitalized with full resumption of normal activities | 1 | Not hospitalized with no limitation of activities |

The percentage of subjects with increasing NIAID score (exhibiting disease progression) and with decreasing NIAID score (exhibiting health improvement) will be presented with the corresponding Clopper-Pearson exact 95% CI, and tested by using Fisher's exact test or Cochran-Mantel-Haenszel test, respectively.

# The percentage of subjects with a negative RT-PCR result for the SARS-CoV-2 (only for SARS-CoV-2 domain) or the influenza virus (only for influenza virus domain) on Day 7

The percentage of subjects with RT-PCR negative results will be tested between treatments by using Chi-square test or Fisher's Exact test.

# Change from baseline in viral load in nasal secretions by RT-PCR (only for SARS-CoV-2 domain)

The viral load and changes in viral load in nasal secretions by RT-PCR will be summarized descriptively by visit. The change from baseline will be analyzed by using ANCOVA.

## Change from baseline in Ct values (only for SARS-CoV-2 domain)

The Ct values and changes in Ct values will be summarized descriptively by visit. The change from baseline will be analyzed by ANCOVA.

#### 7.7.3. Analysis of Exploratory Endpoint

# The percentage of subjects achieving normalized levels on Day 7

Clinical Relevance ("Normal", "Abnormal, non-clinical significant (NCS)" or "Abnormal, clinical

Senhwa Biosciences, Inc. Protocol No.: CX-4945-011 CONFIDENTIAL Version: 3.0/ Date: 16 August, 2024 significant (CS)") of and its transition from baseline will be tabulated descriptively by visit. For subgroup of subjects with baseline levels exceed ULN, Clinical Relevance analyses will be performed additionally, and the percentage of subjects achieving normalized levels on Day 7 will be presented with corresponding Clopper-Pearson exact 95% CI, and tested by using Fisher's exact test or Cochran-Mantel-Haenszel test. Change from baseline in The values and changes in these tests will be summarized descriptively by visit. The change from baseline will be analyzed by using ANCOVA. Note (a): According to the site labs' policy, the or its alternative, the test, will be conducted in the local site labs. To ensure consistency, each site lab should perform the same test

Note (b): If the flow cytometry analyses for are optional at the local site lab.

Changes from baseline in serum cytokine levels: Cytokines to be quantified;

The values and changes in these tests will be summarized descriptively by visit. The change from baseline will be analyzed by using ANCOVA.

# 7.8. Safety Evaluation

All safety assessments, including TEAEs, physical examination, laboratory tests, vital signs, and electrocardiogram results, where indicated, will be presented using descriptive statistics.

# 7.8.1. Treatment-emergent Adverse Events (TEAEs)

throughout the study.

This analysis applies to all treatment-emergent adverse events occurring during the study, recorded in AE eCRF. AEs occurring during the study will be coded using the most recent version of Medical Dictionary for Regulatory Activities (MedDRA). The adverse events will then be grouped by MedDRA preferred terms into frequency tables according to system organ class. All reported adverse events, as well as adverse events judged by the investigator as at least possibly related to IP, will be summarized according to system organ class and preferred term within system organ class. When an adverse event occurs more than once for a subject, the maximal severity to the IP will be counted.

An overview of TEAEs will be presented with number and percentage. Separate summaries will be produced for the following categories, such as TEAEs, SAEs, Treatment-Related TEAEs, TEAEs resulting in discontinuation of study treatment and TEAEs leading to death will be presented. All coding terms will be included in the subject data listing.

#### 7.8.2. Physical Examination

All physical examination findings will be listed. Physical abnormalities will be tabulated descriptively by visit.

## 7.8.3. Laboratory Tests

For continuous data, the values and changes will be summarized descriptively by visit. The change from baseline will be analyzed by using ANCOVA.

For categorical data, the values and transition from baseline will be tabulated descriptively by visit. The transition from baseline will be tested by using Fisher's exact test or Cochran-Mantel-Haenszel test.

Clinical Relevance ("Normal", "Abnormal, non-clinical significant (NCS)" or "Abnormal, clinical significant (CS)") and its transition from baseline will be tabulated descriptively.

#### 7.8.4. Vital Signs

The values and changes in vital signs will be summarized descriptively by visit. The change from baseline will be analyzed by using ANCOVA.

#### 7.8.5. ECG

For overall interpretation, the by visit result and its transition from baseline will be tabulated descriptively by visit. The transition from baseline will be tested by using Fisher's exact test or Cochran-Mantel-Haenszel test.

For continuous data, the values and changes will be summarized descriptively by visit. The change from baseline will be analyzed by using ANCOVA.

# 7.9. Handling of Missing Data

All available data will be displayed and utilized in data analysis. For by-visit efficacy endpoints, ITT analyses applying LOCF (Last Observation Carry Forward) data imputation will be performed additionally as a sensitivity analysis. Refer to Section 7.7.1 ~ 7.7.2 for other missing data estimations. CONFIDENTIAL Version: 3.0/ Date: 16 August, 2024

#### 8. DATA MANAGEMENT

#### 8.1. Data Quality Assurance and Quality Control

Each clinical site will perform internal quality management of study conduct, data and biological specimen collection, documentation and completion.

Quality control (QC) procedures will be implemented on the data entry system and data QC checks that will be run on the database will be generated. Any data or data anomalies will be communicated to the site(s) for clarification/resolution.

Following written Standard Operating Procedures (SOPs), the monitors will verify that the clinical study is conducted and data are generated and biological specimens are collected, documented (recorded), and reported in compliance with the protocol, ICH GCP, and applicable regulatory requirements (e.g., Good Laboratory Practices [GLP], Good Manufacturing Practices [GMP]).

The investigational site will provide direct access to all study-related source data/documents, and reports for the purpose of monitoring and auditing by the sponsor, and inspection by local and regulatory authorities.

#### 8.2. Data Collection and Management Responsibilities

Under the supervision of the site investigator, it is the responsibility of the clinical trial staff at the site to maintain the data collection. The investigator is responsible for ensuring the accuracy, completeness, legibility, and timeliness of the data reported.

Data collection is via Electronic Case Report Form (eCRF) completed by site staff and an electronic Patient Reported Outcome (ePRO) web-based portal by participants. All source documents should be completed in a neat, legible manner to ensure accurate interpretation of data.

Data recorded in the CRF/eCRF derived from source documents should be consistent with the data recorded on the source documents. Study documents should be retained for a period complying with regulations and guidelines applicable to clinical studies of the local countries. No records will be destroyed without the written consent of the sponsor. It is the responsibility of the sponsor to inform the investigator when these documents no longer need to be retained.

Clinical data (including AEs and concomitant medications) and clinical laboratory data will be entered into data capture system, a regulatory authorities compliant data capture system provided by the responsible CRO. The data system includes password protection and internal quality checks, such as automatic range


checks, to identify data that appear inconsistent, incomplete, or inaccurate. Clinical data will be recorded/entered directly from the source documents.


9. DIRECT ACCESS TO SOURCE DATA/DOCUMENTS

9.1. Study Monitoring

Before a study site can enter a patient into the study, a representative of the sponsor will assess the

study site to:

• Determine the adequacy of the facilities

• Discuss with the investigator(s) and other personnel their responsibilities regarding protocol

adherence, and the responsibilities of the sponsor or sponsor's designee. This will be

documented in a separate agreement between the sponsor and the investigator and/or applicable

institution.

During the study, the sponsor or sponsor's designee will have regular contact with the study site for

the following:

• Provide information and support to the investigator(s)

• Confirm that facilities remain acceptable

• Confirm that the investigational team is adhering to the protocol and International Council for

Harmonisation (ICH)/Good Clinical Practice (GCP) guidelines, that data are being accurately

recorded in the CRFs, and that IP accountability checks are being performed

• Perform source data verification. This includes a comparison of the data in the CRFs with the

patient's medical records at the hospital or practice, and other records relevant to the study.

This will require direct access to all original records and/or certified copies for each patient

(e.g., clinic charts).

Record and report any protocol deviations not previously sent to the sponsor

Confirm AEs and SAEs have been properly documented on CRFs and confirm any SAEs have

been forwarded to the sponsor, and those SAEs that met criteria for reporting have been

forwarded to the IRB/IEC

The sponsor or sponsor's designee will be available between visits if the investigator(s) or other staff

needs information or advice.

9.2. Audits and Inspections

Sponsor or sponsor's designee or a designated organization, as well as regulatory authorities and

IRBs/IECs must be permitted to inspect all study-related documents and other materials at the study


site, including the Investigator Site File, the completed CRFs, the IP, and the patients' original medical records/files and/or certified copies. The clinical study protocol, each step of the data capture procedure, and the handling of the data, including the final clinical study report, will be subject to independent Quality Assurance activities. Audits may be conducted at any time during or after the study to ensure the validity and integrity of the study data.

The purpose of a sponsor audit or regulatory inspection is to systematically and independently examine study-related activities and documents to determine whether these activities will be conducted, and data will be recorded, analyzed, and accurately reported according to the protocol, ICH GCP guidelines, and any applicable regulatory requirements. The investigator must contact the sponsor immediately if contacted by a regulatory agency about an inspection.

#### 9.3. Institutional Review Board/Independent Ethics Committee

Prior to the commencement of the study at a given study site, the clinical study protocol will be submitted together with its associated documents (e.g., ICF, patient information sheet, IB, etc.) to the responsible IRB/IEC for its favorable opinion/approval. The written favorable opinion/approval of the IRB/IEC will be filed in the Investigator Site File, and a copy will be filed in the Trial Master File at the sponsor or sponsor's designee.

The study must not start at a study site before the sponsor has obtained written confirmation of favorable opinion/approval from the concerned IRB/IEC. The IRB/IEC will be asked to provide documentation of the date of the meeting at which the favorable opinion/approval will be given, and of the members and voting members present at the meeting. Written evidence of favorable opinion/approval that clearly identifies the study, the clinical study protocol version and the patient information and ICF version reviewed should be provided. Where possible, copies of the meeting minutes should be obtained.

Amendments to the clinical study will also be submitted to the concerned IRB/IEC, before implementation in case of substantial changes. Relevant safety information will be submitted to the IRB/IEC during the study in accordance with national regulations and requirements.

All IRB/IEC approvals and all materials approved by the IRB/IEC for this study including the patient consent form and recruitment materials must be maintained by the Investigator and made available for inspection.

10. ETHICAL AND LEGAL ASPECTS

# Protocol No.: CX-4945-011 CONFIDENTIAL Version: 3.0/ Date: 16 August, 2024

# 10.1. Good Clinical Practice

This study must be carried out in compliance with the protocol and in accordance with sponsor/CRO standard operating procedures. These are designed to ensure adherence to Good Clinical Practice, as described in the following documents:

- 1. ICH Harmonized Tripartite Guidelines for Good Clinical Practice 2016.
- Declaration of Helsinki, concerning medical research in humans (Recommendations Guiding Physicians in Biomedical Research Involving Human Subjects, Helsinki 1964, amended Tokyo 1975, Venice 1983, Hong Kong 1989, Somerset West 1996, Edinburgh, 2000, Washington 2002, Tokyo 2004, Seoul 2008, Fortaleza 2013).

The investigator agrees, when signing the protocol, to adhere to the instructions and procedures described in it and thereby to adhere to the principles of Good Clinical Practice that it conforms to.

#### 10.2. Delegation of Investigator Responsibilities

Responsibilities of the investigators conducting the study in addition to those stated before are enumerated below:

- Obtain Institutional Review Board (IRB) approval to conduct the clinical study.
- Provide the sponsor with written documentation that the study protocol, any protocol amendments, and the informed consent form have received IRB approval.
- Provide the sponsor with a list of IRB members, including their affiliations and qualifications. As
  an alternative, a General Assurance number (as assigned by the Department of Health and Human
  Services) fulfills this requirement.
- Report to the IRB as required. The IRB must assume continued responsibility for the study and review the research on an annual basis.
- Maintain a file of all communications with the IRB on issues related to the clinical trial.
- Conduct the study according to the protocol, ICH GCP guidelines, and in accordance with the Declaration of Helsinki.

#### 10.3. Subject Information and Informed Consent

Written informed consent must be obtained from all subjects prior to study participation. The informed consent form documents the information the investigator provides to the subject and the subject's agreement to participate. The investigator will fully explain the nature of the study, along with the

aims, methods, anticipated benefits, potential hazards, and discomfort that participation might entail.

The informed consent must be signed and dated by each subject or legal representative before entering

the study and prior to the performance of any study specific procedures.

Study site must provide the sponsor (or designee) with a copy of the informed consent approved by

that site's Institutional Review Board (IRB), or Ethics Committee (EC). The subject or the subject's

legally authorized representative must sign the informed consent form. The original signed consent

form will be retained in the subject's study records, and a copy will be provided to the subject. The

sponsor will assure that each informed consent meets the basic elements of informed consent.

10.4. Subject Rights and Confidentiality

10.4.1. Subject confidentiality

The trial staff will ensure that the subjects' anonymity is maintained. The subjects will be identified

only by initials and a subject's ID number on the CRF and any electronic database. All documents will

be stored securely and only accessible by trial staff and authorized personnel. The study will comply

with the local regulation for protecting personal data stored on computers or in an organized paper

filing system which requires data to be anonymized as soon as it is practical to do so.

10.4.2. Study discontinuation

The study may be discontinued at any time by the IRB, FDA/TFDA, or other government agencies as

part of their duties to ensure that research subjects are protected.

10.5. Protocol Amendments

The investigator is responsible for properly notifying the sponsor of protocol changes or revisions. The

investigators without prior written authorization from the sponsor may make no changes to this

protocol.

10.6. Approval of the Study Protocol and Amendments

Before the start of the study, the study protocol, informed consent document, and any other appropriate

documents will be submitted to the independent ethics committee (IEC)/institutional review board

(IRB) with a cover letter or a form listing the documents submitted, their dates of issue, and the site

(or region or area of jurisdiction, as applicable) for which approval is sought. If applicable, the

documents will also be submitted to the authorities, in accordance with local legal requirements.


The IP can only be supplied to the investigator after the sponsor has received documentation on all ethical and legal requirements for starting the study. This documentation must also include a list of the members of the IEC/IRB and their occupations and qualifications. If the IEC/IRB will not disclose the names of the committee members, it should be asked to issue a statement confirming that the composition of the committee is in accordance with GCP. Formal approval by the IEC/IRB should preferably mention the study title, study code, study site (or region or area of jurisdiction, as applicable), and any other documents reviewed. It must mention the date on which the decision is made and must be officially signed by a committee member.

Before the first subject is enrolled in the study, all ethical and legal requirements must be met.

The IEC/IRB and, if applicable, the authorities must be informed of all subsequent protocol amendments, in accordance with local legal requirements. Amendments must be evaluated to determine whether formal approval must be sought and whether the informed consent document should also be revised.

The investigator must keep a record of all communication with the IEC/IRB and, if applicable, between a coordinating investigator and the IEC/IRB. This also applies to any communication between the investigator (or the coordinating investigator, if applicable) and the authorities.

#### 10.7. Publication policy

The sponsor will not suppress or veto publications, but maintains the right to delay publication to ensure against inadvertent disclosure of confidential information or unprotected inventions. Investigators will inform the sponsor in advance of any plans to publish or present data from the study and provide the sponsor an opportunity to review any proposed publication or other type of disclosure before it is submitted or otherwise disclosed. Any publications and presentations of the results (abstracts in journals or newspapers, oral presentations, etc.), either in whole or in part, by investigators or their representatives will require pre-submission review by the sponsor.

Further details regarding the publication of Study results may be described in a separate agreement between the Sponsor and the Investigator and/or applicable institution.


**Protocol Amendment History** Rationale Summary of Change Version Date Initial version 11OCT2023 1.0 NA 2.0 05FEB2024 Revise the primary endpoint Per Sponsor request Revise the secondary endpoints Revise the exploratory endpoints - Revise the inclusion and exclusion criteria - Revise discontinuation of study Intervention - Clarify the concomitant therapy - Clarify Dosage and Administration - Add treatment compliance definition - Revise the period of Visit 1/Screening Visit - Revise the schedule of activity Revise the subject recording platform to ePRO Revise the study assessments - Revise AE and SAE definition and reporting - Add pregnancy reporting - Revise statistical methods Update the abbreviation list Per Sponsor's requests 3.0 16AUG2024 - Add the flow cytometry analyses for CD3 and CD4 - Revise the SOA footnote # 1 and #15 based on NtF No. NTF-C4-011-005 - Clarify the mPP population definition based on NtF No. NTF-C4-011-011 - Add the treatment compliance definition in Section 4.6 - Revise the SOA footnote #4 based on NtF No. NTF-C4-011-003 - Clarify the tests based on NtF No. NTF-

C4-011-006

| Version | Date | Summary of Change | Rationale |
|---------|------|-------------------------------------------------|-----------|
| | | - Revise the exploratory | |
| | | endpoints based on NtF No. | |
| | | NTF-C4-011-008 | |
| | | <ul> <li>Clarify the hospitalization</li> </ul> | |
| | | definition in Sections 5.2.4.1 | |
| | | and 5.2.5.6 based on NtF No. | |
| | | NTF-C4-011-009 | |
| | | - Revise the PP population | |
| | | applied to the safety | |
| | | population | |
| | | - Revise 80 – 120% of 10 | |
| | | doses of the IP for the PP | |
| | | and mPP populations | |
| | | - Add the SOA footnote # 12 | |
| | | for PR-PCR performed in | |
| | | subjects who are early | |
| | | termination | |
| | | - Add the SOA footnote # 18 | |
| | | for one dispensation | |
| | | - Clarify the central or local | |
| | | site lab for performing RT- | |
| | | PCR tests | |
| | | - Update the abbreviation list | |
| | | - Revised some typos | |

#### 11. REFERENCES

- (1) Regunath H, Oba Y. Community-Acquired Pneumonia. 2022 Nov 15. In: StatPearls [Internet]. Treasure Island (FL): StatPearls Publishing; 2023 Jan–.
- (2) Womack J, Kropa J. Community-Acquired Pneumonia in Adults: Rapid Evidence Review. Am Fam Physician. 2022 Jun 1;105(6):625-630.
- (3) Torres A, Cilloniz C, Niederman MS, Menéndez R, Chalmers JD, Wunderink RG, van der Poll T. Pneumonia. Nat Rev Dis Primers. 2021 Apr 8;7(1):25.
- (4) Helena D. Cohen, Rachel W, Julie C, Adam M. Community-acquired pneumonia (non COVID-19), BMJ Best Practice, Last updated: 31 Jan 2023; refer to: https://bestpractice.bmj.com/topics/en-gb/3000108
- (5) Alimi Y, Lim WS, Lansbury L, et al. Systematic review of respiratory viral pathogens identified in adults with community-acquired pneumonia in Europe. J Clin Virol. 2017 Oct;95:26-35.
- (6) Ruuskanen, O., Lahti, E., Jennings, L. C., and Murdoch, D. R. Viral Pneumonia. The Lancet. 2011 377, 1264–1275. doi:10.1016/s0140-6736(10)61459-6
- (7) Andrew M. Freeman; Townes R. Leigh, Jr. Viral Pneumonia. StatPearls [Internet]. Last Update: July 4, 2023; refer to:https://www.ncbi.nlm.nih.gov/books/NBK513286/
- (8) Burk M, El-Kersh K, Saad M, Wiemken T, Ramirez J, Cavallazzi R. Viral infection in community-acquired pneumonia: a systematic review and meta-analysis. Eur Respir Rev. 2016 Jun;25(140):178-88.
- (9) Ren GL, Wang XF, Xu J, Li J, Meng Q, Xie GQ, Huang B, Zhu WC, Lin J, Tang CH, Ye S, Li Z, Zhu J, Tang Z, Ma MX, Xie C, Wu YW, Liu CX, Yang F, Zhou YZ, Zheng Y, Lan SL, Chen JF, Ye F, He Y, Wu BQ, Chen L, Fu SM, Zheng CZ, Shi Y. Comparison of acute pneumonia caused by SARS-COV-2 and other respiratory viruses in children: a retrospective multi-center cohort study during COVID-19 outbreak. Mil Med Res. 2021 Feb 16;8(1):13.
- (10) Attaway AH, Scheraga RG, Bhimraj A, Biehl M, Hatipoğlu U. Severe covid-19 pneumonia: pathogenesis and clinical management. BMJ. 2021 Mar 10;372:n436. doi: 10.1136/bmj.n436. PMID: 33692022.
- (11) Katie Heiser, Peter F. McLean, Chadwick T. Davis, Ben Fogelson, Hannah B. Gordon, Pamela Jacobson, Brett Hurst, Ben Miller, Ronald W. Alfa, Berton A. Earnshaw, Mason L. Victors, Yolanda T. Chong, Imran S. Haque, Adeline S. Low, Christopher C. Gibson. Identification of

- potential treatments for COVID-19 through artificial intelligence-enabled phenomic analysis of human cells infected with SARS-CoV-2, bioRxiv 2020.04.21.054387
- (12) Piirsoo A, Piirsoo M, Kala M, Sankovski E, Lototskaja E, Levin V, et al. (2019) Activity of CK2α protein kinase is required for efficient replication of some HPV types. PLoS Pathog 15(5): e1007788
- (13) Rosenberger, A.F.N., Morrema, T.H.J., Gerritsen, W.H. et al. Increased occurrence of protein kinase CK2 in astrocytes in Alzheimer's disease pathology. J Neuroinflammation 13, 4 (2016).
- (14) Eric Ka-Wai Hui, Debi P. Nayak (2002). Role of G protein and protein kinase signalling in influenza virus budding in MDCK cells. JOURNAL OF GENERAL VIROLOGY, Volume 83, Issue 12
- (15) Koffa MD, Kean J, Zachos G, Rice SA, Clements JB. CK2 protein kinase is stimulated and redistributed by functional herpes simplex virus ICP27 protein. J Virol. 2003;77(7):4315-4325.
- (16) Clinical study report: A Dose Selection Phase 1 Study Evaluating the Safety and Tolerability of Silmitasertib (CX-4945) in Healthy Subjects. Senhwa Biosciences, Inc. [unpublished internal data] 20 June, 2023
- (17) Clinical study report: A Phase II, Randomized and Controlled Investigator Initiated Trial Evaluating Safety, Pharmacokinetics and Clinical Benefit of Silmitasertib (CX-4945) in Outpatient Adult Subjects with Moderate Coronavirus Disease 2019 (COVID-19). Senhwa Biosciences, Inc. [unpublished internal data] 29, September, 2022
- (18) Borad MJ, Bai LY, Richards D, Mody K, Hubbard J, Rha SY, Soong J, McCormick D, Tse E, O'Brien D, Bayat A, Ahn D, Davis SL, Park JO, Oh DY. Silmitasertib plus gemcitabine and cisplatin first-line therapy in locally advanced/metastatic cholangiocarcinoma: A Phase 1b/2 study. Hepatology. 2023 Mar 1;77(3):760-773.
- (19) Rosenberger AF, Morrema TH, Gerritsen WH, van Haastert ES, Snkhchyan H, Hilhorst R, Rozemuller AJ, Scheltens P, van der Vies SM, Hoozemans JJ. Increased occurrence of protein kinase CK2 in astrocytes in Alzheimer's disease pathology. J Neuroinflammation. 2016 Jan 6:13:4.
- (20) de Bourayne M, Gallais Y, El Ali Z, Rousseau P, Damiens MH, Cochet C, Filhol O, Chollet-Martin S, Pallardy M, Kerdine-Römer S. Protein kinase CK2 controls T-cell polarization through dendritic cell activation in response to contact sensitizers. J Leukoc Biol. 2017 Mar;101(3):703-715. doi: 10.1189/jlb.3A0715-320RR. Epub 2016 Oct 5. PMID: 27707883.

